CLINICAL TRIAL: NCT04800211
Title: An Open-Label, Parallel-Group, Controlled Study to Evaluate Changes in Biomarkers of Cigarette Smoke Exposure and Biomarkers of Potential Harm in Adult Smokers Who Completely Switch to Using e-Vapor Products for 24 Weeks
Brief Title: Biomarkers of Exposure and Biomarkers of Potential Harm in Adult Smokers Who Completely Switch to E-vapor Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altria Client Services LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ALCS-RA-16-06/ALCS-RA-17-11-EV
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Intervention Model Description: This research study utilized a parallel-group, open-label, controlled design and was conducted at multiple study sites.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Continue smoking under ad libitum use of subjects' own brand of conventional lit-end cigarettes, without use of any other type of tobacco/nicotine containing product, for the entire duration of study participation.
- Test 1 (Experimental): Exclusive ad libitum use of test e-Vapor Product NuMark LLC, MarkTen® XL Bold CLASSIC* without use of any other type of tobacco/nicotine containing product, for the entire duration of study participation.
  *Product no longer sold commercially
  Interventions: Other: Experimental: Test Product 1
- Test 2 (Experimental): Exclusive ad libitum use of test e-Vapor Product Nu Mark LLC, MarkTen® XL Bold MENTHOL* without use of any other type of tobacco/nicotine containing product, for the entire duration of study participation.
  *Product no longer sold commercially
  Interventions: Other: Experimental: Test Product 2

INTERVENTIONS:
Other: Experimental: Test Product 1 — Subjects were instructed to completely replace their cigarettes with the Test Product 1 EVP (Nu Mark LLC, MarkTen® XL Bold CLASSIC)
  Arms: Test 1
Other: Experimental: Test Product 2 — Subjects were instructed to completely replace their cigarettes with the Test Product 2 EVP (Nu Mark LLC, MarkTen® XL Bold MENTHOL)
  Arms: Test 2

SUMMARY:
The purpose of this study was to estimate changes in biomarkers of exposure (BoE) and biomarkers of potential harm (BoPH) in adult cigarette smokers (AS) who switched to using an e-vapor product (EVP) relative to adult smokers who continue smoking exclusively.

DETAILED DESCRIPTION:
This study was conducted as a randomized, parallel-group, open-label, 24-week, controlled clinical study split into an initial 12-week study (Study 1), with a follow-up at 24 weeks (Study 2) in a sub-population of switchers. For Study 1 a total of 450 subjects were enrolled. Of those subjects who successfully completed Study 1, 150 were then enrolled into Study 2 with no interruption in study participation. The study compared changes in BoE and BoPH in AS who switched to ad libitum use of one of two test EVPs with those in the Control group who continued to smoke conventional cigarettes. The study enrolled AS who were considered to be in overall good health.

ELIGIBILITY:
Inclusion Criteria:

Study 1

Subjects must satisfy the following criteria before being enrolled into the study. Subjects must:

1. sign an IRB-approved informed consent form (ICF) for the study;
2. be between the ages of 30 and 65 years, inclusive, at the time of Screening, Visit 1;
3. have > 500 ng/ml urine cotinine measurement at Screening, Visit 1;
4. have smoked for ≥ 10 years and smoked an average of ≥ 10 manufactured cigarettes per day during the 12 months prior to Screening, Visit 1;

   a) Brief periods [i.e., up to 7 consecutive days] of non smoking during the 12 months prior to Screening, Visit 1 due to illness, trying to quit, or participation in a study where smoking was prohibited are acceptable.
5. indicate that he/she is "definitely" or "probably" willing and able to replace their cigarettes for 12 weeks with the assigned test e-Vapor product;
6. have daily access to text messaging capable cellular phone for daily product use reporting;
7. have a negative ethanol breath test and amphetamines, opiates, cannabinoids, and cocaine urine drug screen results at Screening, Visit 1;

   a) Subjects with a prescription from a licensed physician will not be exempted from this criterion.
8. if female (all females), have a negative serum pregnancy test at Visit 1 and negative urine pregnancy test at Visit 2 through Visit 7, inclusive;
9. if female, heterosexually active, and of childbearing potential (i.e., not surgically sterile or 2 years naturally postmenopausal), must have used a medically accepted method of contraception (listed below in a) and b)) prior to Screening, Visit 1 and must agree to continue to use such method(s) through the End of Study;

   1. Surgically sterile includes bilateral tubal ligation, Essure, hysterectomy, or bilateral oophorectomy at least 6 months prior to Screening, Visit 1. Naturally postmenopausal is defined as women having 2 years without menses.
   2. Acceptable methods of contraception are: hormonal (i.e., oral, transdermal patch, implant, or injection) consistently for at least 3 months prior to Screening, Visit 1; double barrier (i.e., condom with spermicide or diaphragm with spermicide) consistently for at least 4 weeks prior to Screening, Visit 1; and intrauterine device for at least 3 months prior to Screening, Visit 1; or only have a partner who has been vasectomized for at least 6 months prior to Screening, Visit 1.
10. Be willing and able to comply with the requirements of the study.

Study 2

Subjects must satisfy the following criteria before being enrolled into the study. Subject must:

1. have participated in and completed the 12-week ALCS-RA-16-06-EV study and have Baseline biomarker samples collected;
2. demonstrate willingness to participate by signing an Institutional Review Board (IRB)-approved ICF for the study;
3. have demonstrated consistent daily reporting of product use in the 12-week ALCS-RA-16-06-EV (≥ 80% reporting compliance);
4. if randomized to a Test group, have reported an average of no more than 10% of Baseline cigarette smoking per day through Week 11 of the 12-week ALCS-RA-16-06-EV study;
5. if randomized to a Test group, have reported use of at least two Test product cartridges per week in the 12-week ALCS-RA-16-06-EV study;
6. if randomized to a Test group, have exhaled carbon monoxide (eCO) measurements of ≤ 8 ppm at each post-Baseline time point in the 12-week ALCS-RA-16-06-EV study;
7. have daily access to text messaging capable cellular phone for daily product use reporting;
8. if female (all females), have a negative urine pregnancy test at Week 12 (Visit 1) through Week 24 (Visit 5), inclusive;
9. if female, heterosexually active, and of childbearing potential (i.e., not surgically sterile or 2 years naturally postmenopausal), must have used a medically accepted method of contraception (listed below in a) and b)) prior to Screening, Visit 1 of the 12-week ALCS-RA-16-06-EV study and must agree to continue to use such method(s) through Week 24 (EOS);

   1. Surgically sterile includes bilateral tubal ligation, Essure, hysterectomy, or bilateral oophorectomy at least 6 months prior to Screening, Visit 1 of the 12-week ALCS-RA-16-06-EV study. Naturally postmenopausal is defined as women having 2 years without menses.
   2. Acceptable methods of contraception are: hormonal (i.e., oral, transdermal patch, implant, or injection) consistently for at least 3 months prior to Screening, Visit 1 of the 12-week ALCS-RA-16-06-EV study; double barrier (i.e., condom with spermicide or diaphragm with spermicide) consistently for at least 4 weeks prior to Screening, Visit 1 of the 12-week ALCS-RA-16-06-EV study; and intrauterine device for at least 3 months prior to Screening, Visit 1 of the 12-week ALCS-RA-16-06-EV study; or only have a partner who has been vasectomized for at least 6 months prior to Screening, Visit 1 of the 12-week ALCS-RA-16-06-EV study.
10. Be willing and able to comply with the requirements of the study.

Exclusion Criteria:

Study 1

Subjects may be excluded from the study if there is evidence of any of the following criteria. Exceptions may be permitted at the discretion of the Investigator and in consultation with the Sponsor or designee provided there would be no additional risk to the subject. Any exceptions will be documented.

1. History or presence of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, urologic, diabetes, existing respiratory diseases, immunologic, psychiatric, or cardiovascular disease, or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results. (Note: chronic medical conditions controlled and on stable medications [over past 3 months] may not necessarily be exclusionary per Investigator discretion);
2. Currently taking medication for depression, asthma or diabetes;
3. Allergy to menthol;
4. Systolic blood pressure > 140 mmHg and / or diastolic blood pressure > 90 mmHg at Screening Visit 1.
5. Have clinically significant abnormal findings on the physical examination, vital signs, electrocardiogram (ECG), or medical history that would jeopardize the safety of the subject, in the opinion of the Investigator;
6. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV) at Screening, Visit 1;
7. Current evidence or any history of congestive heart failure;
8. Any acute illness (e.g., upper respiratory infection, viral infection) requiring treatment within 2 weeks before Visit 3 (Day 1);
9. History of drug or alcohol abuse within 24 months of Visit 3 (Day 1) as defined by the Investigator;
10. BMI greater than 40.0 kg/m2 or less than 18.0 kg/m2 at Screening, Visit 1;
11. Post-bronchodilator Forced expiratory volume at one second (FEV1):Forced vital capacity (FVC) ratio < 0.7 and FEV1 < 50% of predicted at Screening, Visit 2;
12. Post-bronchodilator FEV1:FVC ratio < 0.75 and FEV1 increase ≥ 12% and > 200 mL from pre- to post-bronchodilator at Screening, Visit 2;
13. Estimated creatinine clearance (by Cockcroft-Gault equation) < 80 mL/min at Screening, Visit 1;
14. Serum alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 1.5 times the upper limit of the reference range at Screening, Visit 1;
15. Female candidates who are pregnant, lactating, or intend to become pregnant from Screening, Visit 1 through End of Study;
16. Use of HDL-C raising medication / supplements (e.g., niacin, gemfibrizole, fenofibrate, etc.) within the past 3 months prior to Screening, Visit 1 or any time during the study;
17. Use of nicotine-containing products other than manufactured cigarettes (e.g., roll-your-own cigarettes, e-cigarette or e-Vapor products, Bidis, snuff, nicotine inhaler, pipe, cigar, smokeless tobacco, nicotine patch, nicotine spray, nicotine lozenge, or nicotine gum) within 14 days prior to Screening, Visit 1 through Visit 3 (Day 1) except as required for the purpose of this study;
18. Donation of blood or blood products, including plasma, history of significant blood loss in the opinion of the investigator, or receipt of whole blood or a blood product transfusion within 60 days prior to Visit 3 (Day 1);
19. Participation in a clinical study of an investigational drug, medical device, biologic, or of a tobacco product, within 30 days before Visit 3 (Day 1);
20. Participation in more than two ALCS studies within 12 months before Visit 3 (Day 1);
21. Already enrolled or failed screening for the current study at a different study site;
22. Subject or a first-degree relative (i.e., parent, spouse, sibling, or child) is a current or former employee of the tobacco industry or a named party or class representative in litigation with any tobacco company.

Study 2

Subjects may be excluded from the study if there is evidence of any of the following. Exceptions may be permitted at the discretion of the Investigator and in consultation with the Sponsor or designee provided there would be no additional risk to the subject. Any exceptions will be documented.

1. Have clinically significant abnormal findings on the physical examination, vital signs, or ECG at the EOS visit (Visit 7) of the 12-week ALCS-RA-16-06-EV study that would jeopardize the safety of the subject, in the opinion of the Investigator;
2. Female subjects who are pregnant (as determined at the EOS visit [Visit 7] of the 12-week study), lactating, or intend to become pregnant from Visit 1 (Week 12) through Week 24 (EOS);
3. Use of any medication for depression, asthma, or diabetes at any time during the study;
4. Use of HDL-C raising medication / supplements (e.g., niacin, gemfibrozil, fenofibrate, etc.) at any time during the study;
5. Subject or a first-degree relative (i.e., parent, spouse, sibling, or child) is a current or former employee of the tobacco industry or a named party or class representative in litigation with any tobacco company;
6. Subject or a first-degree relative (i.e., parent, spouse, sibling, or child) is a current or former employee of Celerion or any of the clinical study sites.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Edmiston, PhD, Study Director — Altria Client Services
Locations (10):
- United States (10):
  - LA Clinical Trials, Burbank, California
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Central Kentucky Research Associates, Lexington, Kentucky
  - DaVita Clinical Research, Minneapolis, Minnesota
  - QPS Bio-Kinetic, Springfield, Missouri
  - Celerion, Lincoln, Nebraska
  - Clinical Research Consortium, Las Vegas, Nevada
  - High Point Clinical Trials Center, High Point, North Carolina
  - Rose Research Center, LLC, Raleigh, North Carolina
  - New Orleans Center for Clinical Research, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After screening, subjects who met all eligibility criteria were randomized to one of the study groups. Eligible subjects who completed ALCS-RA-16-06-EV were entered into the ALCS-RA-17-11-EV 12-week extension study and assigned to the same study groups as the ALCS-RA-16-06-EV study.
Groups:
- Test 1: Exclusive ad libitum use of test e-Vapor Product NuMark LLC, MarkTen® XL Bold CLASSIC* without use of any other type of tobacco/nicotine containing product, for the entire duration of study participation.
  *Product no longer sold commercially
  Experimental: Test Product 1: Subjects were instructed to completely replace their cigarettes with the Test Product 1 EVP (Nu Mark LLC, MarkTen® XL Bold CLASSIC)
- Test 2: Exclusive ad libitum use of test e-Vapor Product Nu Mark LLC, MarkTen® XL Bold MENTHOL* without use of any other type of tobacco/nicotine containing product, for the entire duration of study participation.
  *Product no longer sold commercially
  Experimental: Test Product 2: Subjects were instructed to completely replace their cigarettes with the Test Product 2 EVP (Nu Mark LLC, MarkTen® XL Bold MENTHOL)
Period: ALCS-RA-16-06-EV (Weeks 1-12)
Arm/Group | Test 1 | Test 2 | Control
Started | 151 | 150 | 149
Completed | 121 | 125 | 136
Not Completed | 30 | 25 | 13
Not completed — Adverse Event | 4 | 1 | 0
Not completed — Failure To Meet Ie Post Enrollment | 1 | 0 | 0
Not completed — Lost to Follow-up | 8 | 8 | 2
Not completed — Non-Compliance With Study Procedures | 8 | 7 | 2
Not completed — Other | 1 | 2 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Withdrawal by Subject | 8 | 7 | 5
Period: ALCS-RA-17-11-EV (Weeks 12-24)
Arm/Group | Test 1 | Test 2 | Control
Started | 48 | 50 | 52
Completed | 47 | 50 | 49
Not Completed | 1 | 0 | 3
Not completed — Non-Compliance With Study Procedures | 0 | 0 | 1
Not completed — Other | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Clinical Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Test 1 | Test 2 | Control | Total
Number analyzed (Participants) | 151 | 150 | 149 | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (8.45) | 44.1 (9.26) | 44.4 (10.1) | 44.1 (9.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 75 | 73 | 222
  Male | 77 | 75 | 76 | 228
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 4 | 20
  Not Hispanic or Latino | 143 | 142 | 145 | 430
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 0 | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 44 | 37 | 38 | 119
  White | 103 | 111 | 106 | 320
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 1 | 3
Annual Income [Count of Participants; unit: Participants]
  I DO NOT WISH TO ANSWER | 13 | 17 | 10 | 40
  UNDER $20,000 | 37 | 47 | 45 | 129
  $20,000 - $29,999 | 39 | 25 | 25 | 89
  $30,000 - $39,999 | 25 | 20 | 21 | 66
  $40,000 - $49,999 | 10 | 11 | 12 | 33
  $50,000 - $59,999 | 7 | 8 | 12 | 27
  $60,000 - $74,999 | 5 | 8 | 5 | 18
  $75,000 - $99,000 | 10 | 10 | 9 | 29
  $100,000 - $149,999 | 4 | 4 | 6 | 14
  $150,000 AND OVER | 1 | 0 | 4 | 5
Highest Degree [Count of Participants; unit: Participants]
  I DO NOT WISH TO ANSWER | 0 | 1 | 1 | 2
  GRADES 1 THROUGH 8 (ELEMENTARY) | 1 | 1 | 0 | 2
  GRADES 9 THROUGH 11 (SOME HIGH SCHOOL) | 4 | 9 | 6 | 19
  GRADE 12 OR GED (HIGH SCHOOL GRADUATE) | 61 | 55 | 50 | 166
  COLLEGE 1 YEAR TO 3 YEARS (SOME COLLEGE | 69 | 56 | 66 | 191
  COLLEGE 4 YEARS OR MORE (COLLEGE GRADUATE | 12 | 24 | 19 | 55
  POSTGRADUATE/MASTERS/DOCTORATE/LAW/MD | 3 | 4 | 7 | 14
  OTHER | 1 | 0 | 0 | 1
Weight [Mean (Standard Deviation); unit: kilograms] | 82.0 (17.43) | 82.2 (17.63) | 81.1 (15.90) | 81.8 (16.98)
Body Mass Index [Mean (Standard Deviation); unit: (kg/m²)] | 27.810 (5.1312) | 27.915 (5.1466) | 27.733 (4.9777) | 27.820 (5.0753)
Daily Cigarette Use [Mean (Standard Deviation); unit: Cigarettes per day] — Data was collected from subject responses at screening reporting the number of cigarettes smoked per day (CPD).
  Cigarettes per day | 18.2 (5.71) | 17.0 (5.23) | 17.4 (5.79) | 17.5 (5.59)
Years Smoked [Mean (Standard Deviation); unit: years] | 24.1 (8.32) | 25.0 (9.48) | 24.5 (9.78) | 24.5 (9.20)
Height [Mean (Standard Deviation); unit: cm] | 171.51 (9.402) | 171.40 (9.682) | 171.00 (9.651) | 171.31 (9.560)

OUTCOME MEASURES:

1. Primary Outcome: Summary of Urine Total NNAL and Absolute Change From Baseline (ng/g) by Study Group and Visit From Week 1 to Week 12 (mITT Population) [ALCS-RA-16-06-EV]
Description: Summary of urine total 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) (ng/g) and absolute change from Baseline in Weeks 6 and 12 are presented (Study ALCS-RA-16-06-EV).
  Baseline / Visit 3 (Week 1) = Day 1 Visit 5 (Week 6) = Day 42 ± 3 Visit 7 (Week 12) = Day 84 ± 3
  The first urine void of the day was collected at Visits 3, 5 and 7.
  Urine creatinine concentration was measured in the urine collection and used to adjust the urine biomarker concentration values as follows:
  Urine biomarker (ng/g creatinine) = urine biomarker (pg/mL) x 100 / creatinine (mg/dL)
  Absolute change from baseline = Post Product Use Value - Baseline Value
Time Frame: 12 weeks total with measurement timepoints at Week 1/Baseline, Week 6 and Week 12
Population: Modified Intention-to-Treat (mITT): All subjects were randomized according to the randomization schedule; who used at least one study products after randomization was recorded and for whom there was a valid (within ±3 days of the planned measurement day) baseline and at least one post-baseline biomarker.
Measure: Mean (Standard Deviation); unit: ng/g
Groups:
- Test 1 + Test 2 Group: Combined e-Vapor Use Group
Arm/Group | Test 1 | Test 2 | Test 1 + Test 2 Group | Control
Number analyzed (Participants) | 127 | 131 | 258 | 138
ng/g
  Visit 3 (Baseline): Week 1 | 309.098 (253.5221) | 294.831 (212.1778) | 301.854 (233.0988) | 311.851 (245.2203)
  Visit 5: Week 6: number analyzed (Participants) | 124 | 123 | 247 | 134
  Visit 5: Week 6 | 127.254 (191.0786) | 120.568 (157.7745) | 123.925 (174.9627) | 308.521 (220.7403)
  Visit 7: Week 12: number analyzed (Participants) | 112 | 120 | 232 | 128
  Visit 7: Week 12 | 101.544 (146.4668) | 124.000 (163.0721) | 113.159 (155.3513) | 300.819 (217.6292)
  Change from Baseline (Week 6): number analyzed (Participants) | 124 | 123 | 247 | 134
  Change from Baseline (Week 6) | -180.390 (206.3278) | -173.299 (186.8030) | -176.859 (196.4791) | -8.733 (140.9375)
  Change from Baseline (Week 12): number analyzed (Participants) | 112 | 120 | 232 | 128
  Change from Baseline (Week 12) | -191.327 (220.6982) | -160.201 (192.1456) | -175.228 (206.5607) | -15.898 (149.1447)
Statistical Analysis 1: Comparison: Test 1; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -178.789, 95% CI 2-sided [-204.899 to -152.678] — LSM calculated from the MMRM includes study group, study visit, study group by study visit interaction, gender, age class, BMI class as fixed effects and baseline value as the covariate, with a variance-covariance matrix based on the AIC value
Statistical Analysis 2: Comparison: Test 1; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -184.391, 95% CI 2-sided [-211.184 to -157.598] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 2 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 2 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 2 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 2 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -175.100, 95% CI 2-sided [-200.964 to -149.237] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -161.576, 95% CI 2-sided [-187.543 to -135.609] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Test 1 + Test 2 Group; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 + Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 + Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 + Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 + Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -172.983, 95% CI 2-sided [-192.080 to -153.886] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Control is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Control is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Control is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Control is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p = 0.7781, Mixed Models Analysis; Mean Difference (Net) = -3.585, 95% CI 2-sided [-28.572 to 21.401] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Control is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Control is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Control is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Control is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p = 0.5457, Mixed Models Analysis; Mean Difference (Net) = -7.764, 95% CI 2-sided [-32.993 to 17.465] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -175.203, 95% CI 2-sided [-220.445 to -129.961] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -176.627, 95% CI 2-sided [-222.672 to -130.582] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 2 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 2 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 2 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 2 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -171.515, 95% CI 2-sided [-216.626 to -126.404] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -153.812, 95% CI 2-sided [-199.270 to -108.354] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Test 1 + Test 2 Group vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 + Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 + Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 + Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 + Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -165.220, 95% CI 2-sided [-195.898 to -134.541] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Test 1 vs Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 is equal to Test 2 on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 is NOT equal to Test 2 on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 is equal to Test 2 on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g) in Test 1 is NOT equal to Test 2 on Visit 7 (Week 12). (mITT Population); p = 0.2188, Mixed Models Analysis; Mean Difference (Net) = -22.815, 95% CI 2-sided [-59.223 to 13.593] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Summary of Urine Total NNAL and Absolute Change From Baseline (ng/g) by Study Group and Visit From Week 1 to Week 24 (mITT Population) [ALCS-RA-17-11-EV]
Description: Summary of Urine Total NNAL (ng/g) and absolute change from Baseline in Weeks 12, 18 and 24 are presented (Study ALCS-RA-17-11-EV).
  The first urine void of the day was collected at Visits 1, 3 and 5 of the ALCS-RA-17-11-EV study. Baseline samples were collected Week 1 of the ALCS-RA-16-06-EV study.
  Urine creatinine concentration was measured in the urine collection and used to adjust the urine biomarker concentration value as follows:
  Urine biomarker (ng/g creatinine) = urine biomarker (pg/mL) x 100 / creatinine (mg/dL)
  Change from Baseline was calculated as follows:
  Absolute change from baseline = Post Product Use Value - Baseline Value, where Baseline = values reported on Day 1 (Week 1) of the 12-week ALCS-RA-16-06-EV study
  Baseline = Day 1 (Week 1), Visit 1 = Week 12 (Day 84 ± 3), Visit 3 = Week 18 (Day 126 ± 3), and Visit 5 = Week 24 (Day 168 ± 3), relative to the start of the 12-week ALCS-RA-16-06-EV study
Time Frame: 24 weeks total with measurement timepoints at Week 1/Baseline [ALCS-RA-16-06-EV study]), and Week 12, Week 18 and Week 24 [ALCS-RA-17-11-EV study]
Population: Modified ITT: All subjects were randomized according to the randomization schedule; who used at least one study products after randomization was recorded and for whom there was a valid (within ±3 days of the planned measurement day) baseline and at least one post-baseline biomarker.
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Test 1 | Test 2 | Test 1 + Test 2 Group | Control
Number analyzed (Participants) | 47 | 50 | 97 | 49
ng/g
  Baseline: Week 1 | 258.644 (190.1771) | 294.309 (217.0554) | 277.028 (204.2020) | 368.502 (255.5299)
  Visit 1: Week 12 | 37.240 (74.0723) | 65.631 (105.4324) | 51.875 (92.2293) | 357.472 (261.5709)
  Visit 3: Week 18: number analyzed (Participants) | 40 | 48 | 88 | 47
  Visit 3: Week 18 | 34.715 (73.2359) | 56.986 (110.8673) | 46.863 (95.7548) | 294.906 (194.0554)
  Visit 5: Week 24: number analyzed (Participants) | 42 | 48 | 90 | 44
  Visit 5: Week 24 | 40.991 (80.9328) | 80.808 (174.5894) | 62.227 (139.6906) | 274.912 (186.7002)
  Change from Baseline (Week 12) | -221.403 (177.5875) | -228.678 (187.6797) | -225.153 (181.9443) | -11.030 (130.5603)
  Change from Baseline (Week 18): number analyzed (Participants) | 40 | 48 | 88 | 47
  Change from Baseline (Week 18) | -222.851 (172.2263) | -234.967 (198.3954) | -229.460 (186.0037) | -78.423 (149.1454)
  Change from Baseline (Week 24): number analyzed (Participants) | 42 | 48 | 90 | 44
  Change from Baseline (Week 24) | -218.417 (171.7527) | -215.432 (213.0743) | -216.825 (193.8228) | -85.075 (134.0116)
Statistical Analysis 1: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 1 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 1 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -248.311, 95% CI 2-sided [-286.423 to -210.199] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 1 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 1 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -247.572, 95% CI 2-sided [-280.904 to -214.241] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 1 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 1 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -245.868, 95% CI 2-sided [-284.945 to -206.791] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 2 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 2 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 2 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 2 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -234.942, 95% CI 2-sided [-271.603 to -198.282] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 2 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 2 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 2 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 2 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -244.049, 95% CI 2-sided [-275.269 to -212.829] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -221.385, 95% CI 2-sided [-258.371 to -184.398] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Test 1 + Test 2 Group; Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 1 + Test 2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 1 + Test 2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 1 + Test 2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 1 + Test 2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -233.626, 95% CI 2-sided [-261.113 to -206.140] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Control; Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Control is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Control is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Control is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Control is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.1672, Mixed Models Analysis; Mean Difference (Net) = 26.266, 95% CI 2-sided [-11.130 to 63.661] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Control; Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Control is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Control is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Control is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Control is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0140, Mixed Models Analysis; Mean Difference (Net) = -40.051, 95% CI 2-sided [-71.881 to -8.221] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Control; Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Control is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Control is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Control is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Control is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0288, Mixed Models Analysis; Mean Difference (Net) = -42.635, 95% CI 2-sided [-80.785 to -4.484] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 1 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 1 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -274.577, 95% CI 2-sided [-345.428 to -203.726] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 1 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 1 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -207.521, 95% CI 2-sided [-269.198 to -145.844] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 1 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 1 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -203.233, 95% CI 2-sided [-275.683 to -130.784] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 2 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 2 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -261.208, 95% CI 2-sided [-330.647 to -191.769] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 2 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 2 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -203.998, 95% CI 2-sided [-263.396 to -144.599] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -178.750, 95% CI 2-sided [-249.092 to -108.408] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: Test 1 + Test 2 Group vs Control; Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 1 + Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 1 + Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 1 + Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 1 + Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -190.992, 95% CI 2-sided [-237.134 to -144.850] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: Test 1 vs Test 2; Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 2 is equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 2 is NOT equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Total NNAL (ng/g creatinine) in Test 2 is equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 2 is NOT equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.3590, Mixed Models Analysis; Mean Difference (Net) = -24.483, 95% CI 2-sided [-77.096 to 28.130] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Summary of Whole Blood COHb and Absolute Change From Baseline (% Saturation) by Study Group and Visit From Week 1 to Week 12 (mITT Population) [ALCS-RA-16-06-EV]
Description: Summary of whole blood carboxyhemoglobin (COHb) (% Saturation) and absolute change from Baseline in Weeks 6 and 12 are presented (Study ALCS-RA-16-06-EV).
  Blood samples were collected via direct venipuncture at Visits 3, 5, and 7.
  Absolute change from baseline = Post Product Use Value - Baseline Value
  Baseline / Visit 3 (Week 1) = Day 1 Visit 5 (Week 6) = Day 42 ± 3 Visit 7 (Week 12) = Day 84 ± 3
Time Frame: 12 weeks total with measurement timepoints at Week 1/Baseline, Week 6 and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Test 1 | Test 2 | Test 1 + Test 2 Group | Control
Number analyzed (Participants) | 127 | 131 | 258 | 138
percent saturation
  Visit 3 (Baseline): Week 1 | 5.63 (2.073) | 5.39 (1.868) | 5.51 (1.971) | 5.61 (1.957)
  Visit 5: Week 6: number analyzed (Participants) | 124 | 126 | 250 | 135
  Visit 5: Week 6 | 3.26 (1.790) | 3.10 (1.449) | 3.18 (1.626) | 6.05 (2.029)
  Visit 7: Week 12: number analyzed (Participants) | 111 | 120 | 231 | 128
  Visit 7: Week 12 | 2.99 (1.550) | 2.92 (1.141) | 2.95 (1.351) | 5.68 (1.986)
  Change from Baseline (Week 6): number analyzed (Participants) | 124 | 126 | 250 | 135
  Change from Baseline (Week 6) | -2.34 (2.278) | -2.30 (2.355) | -2.32 (2.313) | 0.40 (1.813)
  Change from Baseline (Week 12): number analyzed (Participants) | 111 | 120 | 231 | 128
  Change from Baseline (Week 12) | -2.49 (2.498) | -2.44 (2.187) | -2.46 (2.337) | 0.07 (1.920)
Statistical Analysis 1: Comparison: Test 1; Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.287, 95% CI 2-sided [-2.582 to -1.992] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 1; Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.415, 95% CI 2-sided [-2.722 to -2.107] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.382, 95% CI 2-sided [-2.673 to -2.090] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.486, 95% CI 2-sided [-2.782 to -2.190] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Test 1 + Test 2 Group; Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 + Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 + Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 + Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 + Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.450, 95% CI 2-sided [-2.668 to -2.233] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Control; Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Control is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Control is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Control is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Control is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p = 0.0012, Mixed Models Analysis; Mean Difference (Net) = 0.466, 95% CI 2-sided [0.185 to 0.747] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Control; Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Control is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Control is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Control is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Control is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p = 0.4957, Mixed Models Analysis; Mean Difference (Net) = 0.099, 95% CI 2-sided [-0.187 to 0.386] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.753, 95% CI 2-sided [-3.266 to -2.239] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.514, 95% CI 2-sided [-3.043 to -1.986] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.848, 95% CI 2-sided [-3.359 to -2.336] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.586, 95% CI 2-sided [-3.105 to -2.066] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Test 1 + Test 2 Group vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 + Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 + Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 + Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 + Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.550, 95% CI 2-sided [-2.901 to -2.199] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Test 1 vs Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is equal to Test 2 on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to Test 2 on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is equal to Test 2 on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to Test 2 on Visit 7 (Week 12). (mITT Population); p = 0.7372, Mixed Models Analysis; Mean Difference (Net) = 0.071, 95% CI 2-sided [-0.346 to 0.489] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Summary of Whole Blood COHb and Absolute Change From Baseline (% Saturation) by Study Group and Visit From Week 1 to Week 24 (mITT Population) [ALCS-RA-17-11-EV]
Description: Summary of Whole Blood COHb (% Saturation) and absolute change from Baseline in Weeks 12, 18 and 24 are presented (Study ALCS-RA-17-11-EV).
  Blood samples were collected via direct venipuncture on Visits 1, 3 and 5 of the ALCS-RA-17-11-EV study. Baseline samples were collected Week 1 of the ALCS-RA-16-06-EV study.
  Change from Baseline was calculated as follows:
  Absolute change from baseline = Post Product Use Value - Baseline Value, where Baseline = values reported on Day 1 (Week 1) of the 12-week ALCS-RA-16-06-EV study
  Baseline = Day 1 (Week 1), Visit 1 = Week 12 (Day 84 ± 3), Visit 3 = Week 18 (Day 126 ± 3), and Visit 5 = Week 24 (Day 168 ± 3), relative to the start of the 12-week ALCS-RA-16-06-EV study
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Test 1 | Test 2 | Test 1 + Test 2 Group | Control
Number analyzed (Participants) | 47 | 50 | 97 | 48
percent saturation
  Baseline: Week 1 | 5.36 (2.096) | 5.27 (1.572) | 5.31 (1.835) | 5.60 (1.607)
  Visit 1: Week 12 | 2.28 (0.786) | 2.52 (0.796) | 2.40 (0.796) | 6.34 (2.052)
  Visit 3: Week 18: number analyzed (Participants) | 39 | 49 | 88 | 46
  Visit 3: Week 18 | 2.61 (0.759) | 2.92 (0.944) | 2.78 (0.876) | 6.74 (1.971)
  Visit 5: Week 24: number analyzed (Participants) | 41 | 47 | 88 | 43
  Visit 5: Week 24 | 2.17 (0.635) | 2.34 (0.940) | 2.26 (0.813) | 5.59 (1.460)
  Change from Baseline (Week 12) | -3.08 (2.252) | -2.75 (1.863) | -2.91 (2.057) | 0.75 (2.019)
  Change from Baseline (Week 18): number analyzed (Participants) | 39 | 49 | 88 | 46
  Change from Baseline (Week 18) | -2.65 (1.940) | -2.33 (1.994) | -2.47 (1.966) | 1.18 (1.894)
  Change from Baseline (Week 24): number analyzed (Participants) | 41 | 47 | 88 | 43
  Change from Baseline (Week 24) | -3.13 (1.947) | -2.89 (1.941) | -3.00 (1.937) | 0.04 (1.511)
Statistical Analysis 1: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 1 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 1 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -3.106, 95% CI 2-sided [-3.502 to -2.710] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 1 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 1 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.824, 95% CI 2-sided [-3.235 to -2.414] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 1 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 1 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -3.228, 95% CI 2-sided [-3.553 to -2.904] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 2 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 2 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.839, 95% CI 2-sided [-3.221 to -2.457] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 2 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 2 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.449, 95% CI 2-sided [-2.828 to -2.070] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -3.023, 95% CI 2-sided [-3.328 to -2.718] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Test 1 + Test 2 Group; Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 1 + Test 2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 + Test 2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 1 + Test 2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 + Test 2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -3.126, 95% CI 2-sided [-3.354 to -2.897] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Control; Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Control is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Control is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Control is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Control is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 0.908, 95% CI 2-sided [0.518 to 1.298] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Control; Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Control is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Control is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Control is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Control is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 1.291, 95% CI 2-sided [0.902 to 1.679] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Control; Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Control is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Control is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Control is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Control is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); p = 0.2772, Mixed Models Analysis; Mean Difference (Net) = 0.174, 95% CI 2-sided [-0.142 to 0.490] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 1 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 1 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -4.014, 95% CI 2-sided [-4.750 to -3.278] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 1 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 1 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -4.115, 95% CI 2-sided [-4.865 to -3.365] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 1 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 1 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -3.403, 95% CI 2-sided [-4.005 to -2.801] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 2 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 2 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -3.747, 95% CI 2-sided [-4.473 to -3.020] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 2 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 2 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -3.740, 95% CI 2-sided [-4.461 to -3.018] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -3.197, 95% CI 2-sided [-3.784 to -2.610] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: Test 1 + Test 2 Group vs Control; Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 1 + Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 + Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 1 + Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 1 + Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -3.300, 95% CI 2-sided [-3.678 to -2.921] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: Test 1 vs Test 2; Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 2 is equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is NOT equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood COHb (% Saturation) in Test 2 is equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood COHb (% Saturation) in Test 2 is NOT equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (MiTT Population); p = 0.3480, Mixed Models Analysis; Mean Difference (Net) = -0.206, 95% CI 2-sided [-0.638 to 0.226] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Summary of Whole Blood WBC Count and Absolute Change From Baseline (10^3 Cells/uL) by Study Group and Visit From Week 1 to Week 12 (mITT Population) [ALCS-RA-16-06-EV]
Description: Summary of whole blood white blood cell (WBC) count (10^3 cells/uL) and absolute change from Baseline in Weeks 6 and 12 are presented (Study ALCS-RA-16-06-EV).
  Blood samples were collected via direct venipuncture at Visits 3, 5, and 7.
  Absolute change from baseline = Post Product Use Value - Baseline Value
  Baseline / Visit 3 (Week 1) = Day 1 Visit 5 (Week 6) = Day 42 ± 3 Visit 7 (Week 12) = Day 84 ± 3
Time Frame: 12 weeks total with measurement timepoints at Week 1/Baseline, Week 6 and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Groups:
- Test 1 + Test 2: Combined e-Vapor Use Group
Arm/Group | Test 1 | Test 2 | Test 1 + Test 2 | Control
Number analyzed (Participants) | 127 | 130 | 257 | 139
10^3 cells/uL
  Visit 3 (Baseline): Week 1 | 7.003 (2.3185) | 6.947 (1.9468) | 6.974 (2.1346) | 6.788 (1.9267)
  Visit 5: Week 6: number analyzed (Participants) | 124 | 125 | 249 | 135
  Visit 5: Week 6 | 6.292 (1.6619) | 6.490 (1.6780) | 6.391 (1.6696) | 6.672 (1.8449)
  Visit 7: Week 12: number analyzed (Participants) | 110 | 119 | 229 | 128
  Visit 7: Week 12 | 6.363 (1.6203) | 6.583 (1.8742) | 6.477 (1.7565) | 6.997 (2.0107)
  Change from Baseline (Week 6): number analyzed (Participants) | 124 | 125 | 249 | 135
  Change from Baseline (Week 6) | -0.656 (1.7850) | -0.490 (1.4902) | -0.573 (1.6424) | -0.098 (1.4878)
  Change from Baseline (Week 12): number analyzed (Participants) | 110 | 119 | 229 | 128
  Change from Baseline (Week 12) | -0.564 (1.8111) | -0.325 (1.8580) | -0.440 (1.8356) | 0.227 (1.6425)
Statistical Analysis 1: Comparison: Test 1; Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 is equal to zero on Visit 5. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to zero on Visit 5. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 is equal to zero on Visit 5. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to zero on Visit 5. (mITT Population); p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -0.716, 95% CI 2-sided [-0.951 to -0.481] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 1; Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 is equal to zero on Visit 7. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to zero on Visit 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 is equal to zero on Visit 7. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to zero on Visit 7. (mITT Population); p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -0.686, 95% CI 2-sided [-0.966 to -0.406] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test 2; Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 2 is equal to zero on Visit 5. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to zero on Visit 5. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 2 is equal to zero on Visit 5. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to zero on Visit 5. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.521, 95% CI 2-sided [-0.755 to -0.288] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Test 2; Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 2 is equal to zero on Visit 7. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to zero on Visit 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 2 is equal to zero on Visit 7. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to zero on Visit 7. (mITT Population); p = 0.0131, Mixed Models Analysis; Mean Difference (Net) = -0.342, 95% CI 2-sided [-0.612 to -0.072] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Test 1 + Test 2; Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 + Test 2 is equal to zero on Visit 7. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 + Test 2 is NOT equal to zero on Visit 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 + Test 2 is equal to zero on Visit 7. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 + Test 2 is NOT equal to zero on Visit 7. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.514, 95% CI 2-sided [-0.712 to -0.316] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Control; Null hypothesis: Whole Blood WBC (x 10^3/uL) in Control is equal to zero on Visit 5. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Control is NOT equal to zero on Visit 5. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood WBC (x 10^3/uL) in Control is equal to zero on Visit 5. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Control is NOT equal to zero on Visit 5. (mITT Population); p = 0.0435, Mixed Models Analysis; Mean Difference (Net) = -0.231, 95% CI 2-sided [-0.455 to -0.007] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Control; Null hypothesis: Whole Blood WBC (x 10^3/uL) in Control is equal to zero on Visit 7. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Control is NOT equal to zero on Visit 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood WBC (x 10^3/uL) in Control is equal to zero on Visit 7. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Control is NOT equal to zero on Visit 7. (mITT Population); p = 0.4012, Mixed Models Analysis; Mean Difference (Net) = 0.111, 95% CI 2-sided [-0.149 to 0.371] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Test 1 vs Control; Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 is equal to Control on Visit 5. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to Control on Visit 5. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 is equal to Control on Visit 5. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to Control on Visit 5. (mITT Population); p = 0.0133, Mixed Models Analysis; Mean Difference (Net) = -0.485, 95% CI 2-sided [-0.895 to -0.074] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Test 1 vs Control; Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 is equal to Control on Visit 7. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to Control on Visit 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 is equal to Control on Visit 7. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to Control on Visit 7. (mITT Population); p = 0.0002, Mixed Models Analysis; Mean Difference (Net) = -0.797, 95% CI 2-sided [-1.277 to -0.317] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Test 2 vs Control; Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 2 is equal to Control on Visit 5. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to Control on Visit 5. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 2 is equal to Control on Visit 5. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to Control on Visit 5. (mITT Population); p = 0.2641, Mixed Models Analysis; Mean Difference (Net) = -0.290, 95% CI 2-sided [-0.699 to 0.119] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Test 2 vs Control; Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 2 is equal to Control on Visit 7. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to Control on Visit 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 2 is equal to Control on Visit 7. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to Control on Visit 7. (mITT Population); p = 0.0639, Mixed Models Analysis; Mean Difference (Net) = -0.453, 95% CI 2-sided [-0.924 to 0.018] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Test 1 + Test 2 vs Control; Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 + Test 2 is equal to Control on Visit 7. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 + Test 2 is NOT equal to Control on Visit 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 + Test 2 is equal to Control on Visit 7. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 + Test 2 is NOT equal to Control on Visit 7. (mITT Population); p = 0.0001, Mixed Models Analysis; Mean Difference (Net) = -0.625, 95% CI 2-sided [-0.945 to -0.305] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Test 1 vs Test 2; Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 is equal to Test 2 on Visit 7. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to Test 2 on Visit 7. (mITT Population); Test type: Equivalence — Null hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 is equal to Test 2 on Visit 7. Alternate hypothesis: Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to Test 2 on Visit 7. (mITT Population); p = 0.0776, Mixed Models Analysis; Mean Difference (Net) = -0.344, 95% CI 2-sided [-0.725 to 0.038] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: Summary of Whole Blood WBC Count and Absolute Change From Baseline (10^3 Cells/uL) by Study Group and Visit From Week 1 to Week 24 (mITT Population) [ALCS-RA-17-11-EV]
Description: Summary of Whole Blood WBC Count (10^3 cells/uL) and absolute change from Baseline in Weeks 12, 18 and 24 are presented (Study ALCS-RA-17-11-EV).
  Blood samples were collected via direct venipuncture on Visits 1, 3 and 5 of the ALCS-RA-17-11-EV study. Baseline samples were collected Week 1 of the ALCS-RA-16-06-EV study.
  Change from Baseline was calculated as follows:
  Absolute change from baseline = Post Product Use Value - Baseline Value, where Baseline = values reported on Day 1 (Week 1) of the 12-week ALCS-RA-16-06-EV study
  Baseline = Day 1 (Week 1), Visit 1 = Week 12 (Day 84 ± 3), Visit 3 = Week 18 (Day 126 ± 3), and Visit 5 = Week 24 (Day 168 ± 3), relative to the start of the 12-week ALCS-RA-16-06-EV study
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Test 1 | Test 2 | Test 1 + Test 2 | Control
Number analyzed (Participants) | 47 | 50 | 97 | 49
10^3 cells/uL
  Baseline: Week 1 | 6.547 (1.6295) | 6.851 (1.8432) | 6.704 (1.7406) | 7.082 (1.9593)
  Visit 1: Week 12: number analyzed (Participants) | 47 | 50 | 97 | 48
  Visit 1: Week 12 | 6.207 (1.6000) | 6.450 (1.7554) | 6.332 (1.6776) | 7.230 (1.9184)
  Visit 3: Week 18: number analyzed (Participants) | 40 | 49 | 89 | 47
  Visit 3: Week 18 | 5.986 (1.2707) | 6.642 (1.7254) | 6.347 (1.5643) | 7.073 (2.0805)
  Visit 5: Week 24: number analyzed (Participants) | 42 | 47 | 89 | 44
  Visit 5: Week 24 | 5.972 (1.2750) | 6.152 (1.4051) | 6.067 (1.3408) | 7.401 (1.6116)
  Change from Baseline (Week 12): number analyzed (Participants) | 47 | 50 | 97 | 48
  Change from Baseline (Week 12) | -0.340 (1.3015) | -0.402 (1.7483) | -0.372 (1.5404) | 0.174 (1.9309)
  Change from Baseline (Week 18): number analyzed (Participants) | 40 | 49 | 89 | 47
  Change from Baseline (Week 18) | -0.521 (1.2722) | -0.224 (1.9141) | -0.357 (1.6547) | 0.035 (1.9567)
  Change from Baseline (Week 24): number analyzed (Participants) | 42 | 47 | 89 | 44
  Change from Baseline (Week 24) | -0.622 (1.5029) | -0.762 (1.5132) | -0.696 (1.5014) | 0.202 (1.5842)
Statistical Analysis 1: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 1 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 1 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0055, Mixed Models Analysis; Mean Difference (Net) = -0.621, 95% CI 2-sided [-1.055 to -0.186] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 1 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 1 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0011, Mixed Models Analysis; Mean Difference (Net) = -0.778, 95% CI 2-sided [-1.240 to -0.316] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 1 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 1 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.900, 95% CI 2-sided [-1.260 to -0.540] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 2 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 2 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0150, Mixed Models Analysis; Mean Difference (Net) = -0.520, 95% CI 2-sided [-0.938 to -0.103] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 2 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 2 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.1048, Mixed Models Analysis; Mean Difference (Net) = -0.349, 95% CI 2-sided [-0.771 to 0.074] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.846, 95% CI 2-sided [-1.185 to -0.507] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Test 1 + Test 2; Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 1 + Test 2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 1 + Test 2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 1 + Test 2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 1 + Test 2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.873, 95% CI 2-sided [-1.127 to -0.619] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Control; Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Control is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Control is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Control is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Control is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.2525, Mixed Models Analysis; Mean Difference (Net) = 0.247, 95% CI 2-sided [-0.178 to 0.671] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Control; Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Control is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Control is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Control is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Control is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.6503, Mixed Models Analysis; Mean Difference (Net) = 0.098, 95% CI 2-sided [-0.330 to 0.527] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Control; Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Control is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Control is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Control is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Control is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.1759, Mixed Models Analysis; Mean Difference (Net) = 0.239, 95% CI 2-sided [-0.109 to 0.588] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 1 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 1 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0293, Mixed Models Analysis; Mean Difference (Net) = -0.867, 95% CI 2-sided [-1.674 to -0.060] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 1 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 1 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0362, Mixed Models Analysis; Mean Difference (Net) = -0.876, 95% CI 2-sided [-1.714 to -0.038] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 1 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 1 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.139, 95% CI 2-sided [-1.809 to -0.469] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 2 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 2 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0621, Mixed Models Analysis; Mean Difference (Net) = -0.767, 95% CI 2-sided [-1.559 to 0.025] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 2 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 2 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.5259, Mixed Models Analysis; Mean Difference (Net) = -0.447, 95% CI 2-sided [-1.246 to 0.352] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.085, 95% CI 2-sided [-1.736 to -0.435] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: Test 1 + Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 1 + Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 1 + Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 1 + Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 1 + Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -1.112, 95% CI 2-sided [-1.532 to -0.693] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: Test 1 vs Test 2; Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 2 is equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Whole Blood WBC (x 10^3/uL) in Test 2 is equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.8248, Mixed Models Analysis; Mean Difference (Net) = -0.054, 95% CI 2-sided [-0.535 to 0.427] — [estimate comment as in outcome 1, analysis 1]

7. Primary Outcome: Summary of Serum HDL-C and Absolute Change From Baseline (mg/dL) by Study Group and Visit From Week 1 to Week 12 (mITT Population) [ALCS-RA-16-06-EV]
Description: Summary of serum high density lipoprotein cholesterol (HDL-C) (mg/dL) and absolute change from Baseline in Weeks 6 and 12 are presented (Study ALCS-RA-16-06-EV).
  Blood samples were collected via direct venipuncture at Visits 3, 5, and 7.
  Absolute change from baseline = Post Product Use Value - Baseline Value
  Baseline / Visit 3 (Week 1) = Day 1 Visit 5 (Week 6) = Day 42 ± 3 Visit 7 (Week 12) = Day 84 ± 3
Time Frame: 12 weeks total with measurement timepoints at Week 1/Baseline, Week 6 and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Test 1 | Test 2 | Test 1 + Test 2 | Control
Number analyzed (Participants) | 125 | 130 | 255 | 138
mg/dL
  Visit 3 (Baseline): Week 1 | 44.8 (14.15) | 46.1 (12.56) | 45.5 (13.35) | 46.8 (16.84)
  Visit 5: Week 6: number analyzed (Participants) | 122 | 125 | 247 | 135
  Visit 5: Week 6 | 47.2 (15.01) | 48.0 (12.52) | 47.6 (13.78) | 47.6 (18.13)
  Visit 7: Week 12: number analyzed (Participants) | 110 | 119 | 229 | 128
  Visit 7: Week 12 | 47.3 (14.43) | 48.9 (14.52) | 48.2 (14.46) | 47.4 (18.00)
  Change from Baseline (Week 6): number analyzed (Participants) | 122 | 125 | 247 | 135
  Change from Baseline (Week 6) | 2.3 (6.15) | 1.6 (7.47) | 2.0 (6.84) | 0.6 (10.36)
  Change from Baseline (Week 12): number analyzed (Participants) | 110 | 119 | 229 | 128
  Change from Baseline (Week 12) | 3.3 (6.68) | 3.1 (9.37) | 3.2 (8.17) | 0.8 (8.88)
Statistical Analysis 1: Comparison: Test 1; Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p = 0.0002, Mixed Models Analysis; Mean Difference (Net) = 2.821, 95% CI 2-sided [1.369 to 4.273] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 1; Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.468, 95% CI 2-sided [1.850 to 5.086] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p = 0.0022, Mixed Models Analysis; Mean Difference (Net) = 2.245, 95% CI 2-sided [0.812 to 3.679] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.329, 95% CI 2-sided [1.768 to 4.891] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Test 1 + Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 + Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 + Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 + Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 + Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 3.399, 95% CI 2-sided [2.252 to 4.545] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Control; Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Control is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Control is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Control is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Control is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p = 0.0761, Mixed Models Analysis; Mean Difference (Net) = 1.250, 95% CI 2-sided [-0.132 to 2.633] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Control; Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Control is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Control is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Control is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Control is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p = 0.0211, Mixed Models Analysis; Mean Difference (Net) = 1.778, 95% CI 2-sided [0.269 to 3.286] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); p = 0.3841, Mixed Models Analysis; Mean Difference (Net) = 1.570, 95% CI 2-sided [-0.951 to 4.092] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p = 0.3934, Mixed Models Analysis; Mean Difference (Net) = 1.690, 95% CI 2-sided [-1.084 to 4.464] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); p = 0.7782, Mixed Models Analysis; Mean Difference (Net) = 0.995, 95% CI 2-sided [-1.505 to 3.494] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p = 0.4576, Mixed Models Analysis; Mean Difference (Net) = 1.552, 95% CI 2-sided [-1.171 to 4.274] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Test 1 + Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 + Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 + Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 + Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 + Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p = 0.0849, Mixed Models Analysis; Mean Difference (Net) = 1.621, 95% CI 2-sided [-0.224 to 3.466] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Test 1 vs Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is equal to Test 2 on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to Test 2 on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is equal to Test 2 on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to Test 2 on Visit 7 (Week 12). (mITT Population); p = 0.9016, Mixed Models Analysis; Mean Difference (Net) = 0.139, 95% CI 2-sided [-2.064 to 2.341] — [estimate comment as in outcome 1, analysis 1]

8. Primary Outcome: Summary of Serum HDL-C and Absolute Change From Baseline (mg/dL) by Study Group and Visit From Week 1 to Week 24 (mITT Population) [ALCS-RA-17-11-EV]
Description: Summary of serum HDL-C (mg/dL) and absolute change from Baseline in Weeks 12, 18 and 24 are presented (Study ALCS-RA-17-11-EV).
  Blood samples were collected via direct venipuncture on Visits 1, 3 and 5 of the ALCS-RA-17-11-EV study. Baseline samples were collected Week 1 of the ALCS-RA-16-06-EV study.
  Change from Baseline was calculated as follows:
  Absolute change from baseline = Post Product Use Value - Baseline Value, where Baseline = values reported on Day 1 (Week 1) of the 12-week ALCS-RA-16-06-EV study
  Baseline = Day 1 (Week 1), Visit 1 = Week 12 (Day 84 ± 3), Visit 3 = Week 18 (Day 126 ± 3), and Visit 5 = Week 24 (Day 168 ± 3), relative to the start of the 12-week ALCS-RA-16-06-EV study
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Test 1 | Test 2 | Test 1 + Test 2 | Control
Number analyzed (Participants) | 46 | 49 | 95 | 49
mg/dL
  Baseline: Week 1 | 46.3 (13.05) | 45.2 (12.29) | 45.7 (12.61) | 44.4 (16.04)
  Visit 1: Week 12 | 50.4 (14.44) | 50.7 (16.02) | 50.5 (15.19) | 44.0 (21.54)
  Visit 3: Week 18: number analyzed (Participants) | 39 | 48 | 87 | 47
  Visit 3: Week 18 | 48.4 (13.35) | 47.8 (14.61) | 48.1 (13.98) | 44.0 (22.75)
  Visit 5: Week 24: number analyzed (Participants) | 41 | 46 | 87 | 44
  Visit 5: Week 24 | 50.6 (17.37) | 48.5 (17.95) | 49.5 (17.61) | 40.8 (13.01)
  Change from Baseline (Week 12) | 4.2 (6.51) | 5.5 (11.96) | 4.8 (9.68) | -0.4 (10.10)
  Change from Baseline (Week 18): number analyzed (Participants) | 39 | 48 | 87 | 47
  Change from Baseline (Week 18) | 1.5 (5.80) | 2.8 (12.20) | 2.2 (9.83) | -0.2 (12.26)
  Change from Baseline (Week 24): number analyzed (Participants) | 41 | 46 | 87 | 44
  Change from Baseline (Week 24) | 4.1 (9.02) | 3.5 (13.67) | 3.8 (11.65) | -1.1 (6.79)
Statistical Analysis 1: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 1 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 1 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0004, Mixed Models Analysis; Mean Difference (Net) = 5.587, 95% CI 2-sided [2.511 to 8.662] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 1 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 1 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.1141, Mixed Models Analysis; Mean Difference (Net) = 2.556, 95% CI 2-sided [-0.620 to 5.732] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 1 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 1 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0007, Mixed Models Analysis; Mean Difference (Net) = 5.536, 95% CI 2-sided [2.367 to 8.705] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 2 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 2 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 6.629, 95% CI 2-sided [3.680 to 9.577] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 2 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 2 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0072, Mixed Models Analysis; Mean Difference (Net) = 4.083, 95% CI 2-sided [1.118 to 7.047] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0023, Mixed Models Analysis; Mean Difference (Net) = 4.688, 95% CI 2-sided [1.691 to 7.686] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Test 1 + Test 2; Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 1 + Test 2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 + Test 2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 1 + Test 2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 + Test 2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = 5.112, 95% CI 2-sided [2.874 to 7.350] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Control; Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Control is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Control is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Control is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Control is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.6030, Mixed Models Analysis; Mean Difference (Net) = 0.777, 95% CI 2-sided [-2.165 to 3.720] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Control; Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Control is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Control is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Control is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Control is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.5053, Mixed Models Analysis; Mean Difference (Net) = 1.003, 95% CI 2-sided [-1.960 to 3.967] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Control; Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Control is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Control is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Control is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Control is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.6607, Mixed Models Analysis; Mean Difference (Net) = 0.674, 95% CI 2-sided [-2.347 to 3.694] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 1 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 1 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.1309, Mixed Models Analysis; Mean Difference (Net) = 4.809, 95% CI 2-sided [-0.827 to 10.446] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 1 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 1 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.9776, Mixed Models Analysis; Mean Difference (Net) = 1.553, 95% CI 2-sided [-4.212 to 7.318] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 1 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 1 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.1422, Mixed Models Analysis; Mean Difference (Net) = 4.862, 95% CI 2-sided [-0.939 to 10.663] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 2 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 2 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0334, Mixed Models Analysis; Mean Difference (Net) = 5.851, 95% CI 2-sided [0.307 to 11.396] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 2 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 2 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.5622, Mixed Models Analysis; Mean Difference (Net) = 3.080, 95% CI 2-sided [-2.501 to 8.660] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.2841, Mixed Models Analysis; Mean Difference (Net) = 4.014, 95% CI 2-sided [-1.643 to 9.672] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: Test 1 + Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 1 + Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 + Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 1 + Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 + Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0178, Mixed Models Analysis; Mean Difference (Net) = 4.438, 95% CI 2-sided [0.774 to 8.103] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: Test 1 vs Test 2; Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 2 is equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is NOT equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Serum HDL-C (mg/dL) in Test 2 is equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 2 is NOT equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.6944, Mixed Models Analysis; Mean Difference (Net) = 0.847, 95% CI 2-sided [-3.398 to 5.093] — [estimate comment as in outcome 1, analysis 1]

9. Primary Outcome: Summary of Urine 8-epi-prostaglandin F2alpha and Absolute Change From Baseline (ng/g) by Study Group and Visit From Week 1 to Week 12 (mITT Population) [ALCS-RA-16-06-EV]
Description: Summary of urine 8-epi-prostaglandin F2alpha (ng/g) and absolute change from Baseline in Weeks 6 and 12 are presented (Study ALCS-RA-16-06-EV).
  Baseline / Visit 3 (Week 1) = Day 1 Visit 5 (Week 6) = Day 42 ± 3 Visit 7 (Week 12) = Day 84 ± 3
  The first urine void of the day was collected at Visits 3, 5 and 7.
  Urine creatinine concentration was measured in the urine collection and used to adjust the urine biomarker concentration values as follows:
  Urine biomarker (ng/g creatinine) = urine biomarker (pg/mL) x 100 / creatinine (mg/dL)
  Absolute change from baseline = Post Product Use Value - Baseline Value
Time Frame: 12 weeks total with measurement timepoints at Week 1/Baseline, Week 6 and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Test 1 | Test 2 | Test 1 + Test 2 | Control
Number analyzed (Participants) | 127 | 131 | 258 | 138
ng/g
  Visit 3 (Baseline): Week 1 | 377.138 (211.0106) | 355.984 (177.9443) | 366.397 (194.8302) | 368.710 (200.0174)
  Visit 5: Week 6: number analyzed (Participants) | 124 | 122 | 246 | 134
  Visit 5: Week 6 | 332.952 (212.6164) | 315.095 (150.5924) | 324.096 (184.3240) | 346.856 (195.7020)
  Visit 7: Week 12: number analyzed (Participants) | 111 | 120 | 231 | 128
  Visit 7: Week 12 | 332.455 (219.2878) | 335.687 (143.1724) | 334.134 (183.3207) | 355.639 (233.4254)
  Change from Baseline (Week 6): number analyzed (Participants) | 124 | 122 | 246 | 134
  Change from Baseline (Week 6) | -44.354 (162.5679) | -33.320 (120.3646) | -38.882 (143.0167) | -15.247 (141.7366)
  Change from Baseline (Week 12): number analyzed (Participants) | 111 | 120 | 231 | 128
  Change from Baseline (Week 12) | -39.547 (191.4551) | -18.092 (135.9049) | -28.401 (164.9314) | -7.204 (178.4608)
Statistical Analysis 1: Comparison: Test 1; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p = 0.0031, Mixed Models Analysis; Mean Difference (Net) = -35.556, 95% CI 2-sided [-59.038 to -12.075] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 1; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p = 0.0371, Mixed Models Analysis; Mean Difference (Net) = -31.350, 95% CI 2-sided [-60.818 to -1.882] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p = 0.0043, Mixed Models Analysis; Mean Difference (Net) = -34.356, 95% CI 2-sided [-57.877 to -10.834] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p = 0.2091, Mixed Models Analysis; Mean Difference (Net) = -18.096, 95% CI 2-sided [-46.375 to 10.183] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Test 1 + Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 + Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 + Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 + Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 + Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p = 0.0197, Mixed Models Analysis; Mean Difference (Net) = -24.723, 95% CI 2-sided [-45.473 to -3.973] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Control is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Control is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Control is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Control is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p = 0.2353, Mixed Models Analysis; Mean Difference (Net) = -13.595, 95% CI 2-sided [-36.080 to 8.891] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Control is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Control is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Control is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Control is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p = 0.7329, Mixed Models Analysis; Mean Difference (Net) = -4.759, 95% CI 2-sided [-32.159 to 22.641] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); p = 0.5420, Mixed Models Analysis; Mean Difference (Net) = -21.962, 95% CI 2-sided [-62.989 to 19.065] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p = 0.5234, Mixed Models Analysis; Mean Difference (Net) = -26.591, 95% CI 2-sided [-77.049 to 23.866] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); p = 0.5975, Mixed Models Analysis; Mean Difference (Net) = -20.761, 95% CI 2-sided [-61.867 to 20.344] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p = 0.9331, Mixed Models Analysis; Mean Difference (Net) = -13.337, 95% CI 2-sided [-62.853 to 36.179] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Test 1 + Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 + Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 + Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 + Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 + Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p = 0.2444, Mixed Models Analysis; Mean Difference (Net) = -19.964, 95% CI 2-sided [-53.637 to 13.709] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Test 1 vs Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to Test 2 on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to Test 2 on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to Test 2 on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to Test 2 on Visit 7 (Week 12). (mITT Population); p = 0.5169, Mixed Models Analysis; Mean Difference (Net) = -13.254, 95% CI 2-sided [-53.427 to 26.919] — [estimate comment as in outcome 1, analysis 1]

10. Primary Outcome: Summary of Urine 8-epi-prostaglandin F2alpha and Absolute Change From Baseline (ng/g) by Study Group and Visit From Week 1 to Week 24 (mITT Population) [ALCS-RA-17-11-EV]
Description: Summary of urine 8-epi-prostaglandin F2alpha (ng/g) and absolute change from Baseline in Weeks 12, 18 and 24 are presented (Study ALCS-RA-17-11-EV).
  The first urine void of the day was collected at Visits 1, 3 and 5 of the ALCS-RA-17-11-EV study. Baseline samples were collected Week 1 of the ALCS-RA-16-06-EV study.
  Urine creatinine concentration was measured in the urine collection and used to adjust the urine biomarker concentration value as follows:
  Urine biomarker (ng/g creatinine) = urine biomarker (pg/mL) x 100 / creatinine (mg/dL)
  Change from Baseline was calculated as follows:
  Absolute change from baseline = Post Product Use Value - Baseline Value, where Baseline = values reported on Day 1 (Week 1) of the 12-week ALCS-RA-16-06-EV study
  Baseline = Day 1 (Week 1), Visit 1 = Week 12 (Day 84 ± 3), Visit 3 = Week 18 (Day 126 ± 3), and Visit 5 = Week 24 (Day 168 ± 3), relative to the start of the 12-week ALCS-RA-16-06-EV study
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Test 1 | Test 2 | Test 1 + Test 2 | Control
Number analyzed (Participants) | 47 | 50 | 97 | 49
ng/g
  Baseline: Week 1 | 331.217 (145.3767) | 359.269 (204.4360) | 345.677 (177.9266) | 421.529 (277.7803)
  Visit 1: Week 12: number analyzed (Participants) | 46 | 50 | 96 | 49
  Visit 1: Week 12 | 295.921 (199.4031) | 337.996 (138.6722) | 317.835 (170.8786) | 413.638 (328.9100)
  Visit 3: Week 18: number analyzed (Participants) | 40 | 48 | 88 | 47
  Visit 3: Week 18 | 251.448 (105.3359) | 314.650 (145.3787) | 285.922 (131.8840) | 403.656 (359.5415)
  Visit 5: Week 24: number analyzed (Participants) | 42 | 48 | 90 | 44
  Visit 5: Week 24 | 305.481 (310.8112) | 331.678 (190.5315) | 319.453 (252.6784) | 344.100 (142.3191)
  Change from Baseline (Week 12): number analyzed (Participants) | 46 | 50 | 96 | 49
  Change from Baseline (Week 12) | -35.569 (162.6996) | -21.273 (159.7813) | -28.123 (160.4950) | -7.891 (226.9262)
  Change from Baseline (Week 18): number analyzed (Participants) | 40 | 48 | 88 | 47
  Change from Baseline (Week 18) | -87.745 (92.1074) | -48.891 (115.7881) | -66.552 (106.8853) | -20.874 (255.5397)
  Change from Baseline (Week 24): number analyzed (Participants) | 42 | 48 | 90 | 44
  Change from Baseline (Week 24) | -32.869 (328.5303) | -31.868 (179.4879) | -32.335 (258.3306) | -54.946 (159.6202)
Statistical Analysis 1: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.1359, Mixed Models Analysis; Mean Difference (Net) = -40.174, 95% CI 2-sided [-93.120 to 12.772] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0129, Mixed Models Analysis; Mean Difference (Net) = -71.725, 95% CI 2-sided [-127.961 to -15.490] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.3262, Mixed Models Analysis; Mean Difference (Net) = -37.308, 95% CI 2-sided [-112.293 to 37.678] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.4343, Mixed Models Analysis; Mean Difference (Net) = -20.012, 95% CI 2-sided [-70.468 to 30.444] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0967, Mixed Models Analysis; Mean Difference (Net) = -44.657, 95% CI 2-sided [-97.481 to 8.167] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.4198, Mixed Models Analysis; Mean Difference (Net) = -28.974, 95% CI 2-sided [-99.915 to 41.966] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Test 1 + Test 2; Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 + Test 2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 + Test 2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 + Test 2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 + Test 2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.2121, Mixed Models Analysis; Mean Difference (Net) = -33.141, 95% CI 2-sided [-85.475 to 19.193] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Control; Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Control is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Control is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Control is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Control is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.5445, Mixed Models Analysis; Mean Difference (Net) = 15.799, 95% CI 2-sided [-35.614 to 67.212] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Control; Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Control is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Control is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Control is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Control is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.9534, Mixed Models Analysis; Mean Difference (Net) = 1.583, 95% CI 2-sided [-51.951 to 55.116] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Control; Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Control is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Control is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Control is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Control is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.8366, Mixed Models Analysis; Mean Difference (Net) = 7.584, 95% CI 2-sided [-65.126 to 80.295] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.5437, Mixed Models Analysis; Mean Difference (Net) = -55.973, 95% CI 2-sided [-154.862 to 42.916] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.2974, Mixed Models Analysis; Mean Difference (Net) = -73.308, 95% CI 2-sided [-177.224 to 30.608] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.9026, Mixed Models Analysis; Mean Difference (Net) = -44.892, 95% CI 2-sided [-181.909 to 92.126] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.8954, Mixed Models Analysis; Mean Difference (Net) = -35.811, 95% CI 2-sided [-132.513 to 60.891] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.7485, Mixed Models Analysis; Mean Difference (Net) = -46.239, 95% CI 2-sided [-146.766 to 54.288] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.9578, Mixed Models Analysis; Mean Difference (Net) = -36.559, 95% CI 2-sided [-169.770 to 96.653] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: Test 1 + Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 + Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 + Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 + Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 1 + Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.3635, Mixed Models Analysis; Mean Difference (Net) = -40.725, 95% CI 2-sided [-129.208 to 47.757] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: Test 1 vs Test 2; Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is NOT equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 8-epi-prostaglandin F2alpha (ng/g creatinine) in Test 2 is NOT equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.8713, Mixed Models Analysis; Mean Difference (Net) = -8.333, 95% CI 2-sided [-110.097 to 93.431] — [estimate comment as in outcome 1, analysis 1]

11. Primary Outcome: Summary of Urine 11-dehydrothromboxane B2 and Absolute Change From Baseline (ng/g) by Study Group and Visit From Week 1 to Week 12 (mITT Population) [ALCS-RA-16-06-EV]
Description: Summary of urine 11-dehydrothromboxane B2 (ng/g) and absolute change from Baseline in Weeks 6 and 12 are presented (Study ALCS-RA-16-06-EV).
  Baseline / Visit 3 (Week 1) = Day 1 Visit 5 (Week 6) = Day 42 ± 3 Visit 7 (Week 12) = Day 84 ± 3
  The first urine void of the day was collected at Visits 3, 5 and 7.
  Urine creatinine concentration was measured in the urine collection and used to adjust the urine biomarker concentration values as follows:
  Urine biomarker (ng/g creatinine) = urine biomarker (pg/mL) x 100 / creatinine (mg/dL)
  Absolute change from baseline = Post Product Use Value - Baseline Value
Time Frame: 12 weeks total with measurement timepoints at Week 1/Baseline, Week 6 and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Test 1 | Test 2 | Test 1 + Test 2 Group | Control
Number analyzed (Participants) | 126 | 131 | 257 | 136
ng/g
  Visit 3 (Baseline): Week 1 | 824.877 (726.5075) | 761.598 (518.6039) | 792.622 (628.7305) | 785.424 (457.4472)
  Visit 5: Week 6: number analyzed (Participants) | 123 | 122 | 245 | 132
  Visit 5: Week 6 | 680.700 (371.6959) | 614.562 (312.1994) | 647.766 (344.2553) | 776.000 (480.7616)
  Visit 7: Week 12: number analyzed (Participants) | 110 | 120 | 230 | 125
  Visit 7: Week 12 | 703.664 (444.1672) | 714.007 (413.0628) | 709.060 (427.3102) | 777.506 (471.4327)
  Change from Baseline (Week 6): number analyzed (Participants) | 123 | 122 | 245 | 132
  Change from Baseline (Week 6) | -148.001 (660.1311) | -141.502 (409.6231) | -144.765 (548.7304) | -2.414 (427.2816)
  Change from Baseline (Week 12): number analyzed (Participants) | 110 | 120 | 230 | 125
  Change from Baseline (Week 12) | -47.736 (488.1213) | -55.751 (486.6897) | -51.917 (486.3259) | 5.028 (424.6884)
Statistical Analysis 1: Comparison: Test 1; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p = 0.0003, Mixed Models Analysis; Mean Difference (Net) = -115.256, 95% CI 2-sided [-177.973 to -52.539] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 1; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p = 0.0467, Mixed Models Analysis; Mean Difference (Net) = -74.904, 95% CI 2-sided [-148.706 to -1.102] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -144.035, 95% CI 2-sided [-206.668 to -81.402] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p = 0.0807, Mixed Models Analysis; Mean Difference (Net) = -62.755, 95% CI 2-sided [-133.221 to 7.710] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Test 1 + Test 2 Group; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 + Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 + Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 + Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 + Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p = 0.0095, Mixed Models Analysis; Mean Difference (Net) = -68.830, 95% CI 2-sided [-120.753 to -16.907] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Control is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Control is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Control is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Control is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p = 0.9586, Mixed Models Analysis; Mean Difference (Net) = -1.593, 95% CI 2-sided [-61.873 to 58.687] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Control is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Control is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Control is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Control is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p = 0.9402, Mixed Models Analysis; Mean Difference (Net) = -2.635, 95% CI 2-sided [-71.714 to 66.443] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); p = 0.0390, Mixed Models Analysis; Mean Difference (Net) = -113.663, 95% CI 2-sided [-223.330 to -3.996] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p = 0.4543, Mixed Models Analysis; Mean Difference (Net) = -72.269, 95% CI 2-sided [-199.091 to 54.554] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); p = 0.0051, Mixed Models Analysis; Mean Difference (Net) = -142.442, 95% CI 2-sided [-252.080 to -32.805] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p = 0.6061, Mixed Models Analysis; Mean Difference (Net) = -60.120, 95% CI 2-sided [-184.286 to 64.046] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Test 1 + Test 2 Group vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 + Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 + Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 + Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 + Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p = 0.1242, Mixed Models Analysis; Mean Difference (Net) = -66.194, 95% CI 2-sided [-150.672 to 18.284] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Test 1 vs Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to Test 2 on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to Test 2 on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to Test 2 on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to Test 2 on Visit 7 (Week 12). (mITT Population); p = 0.8117, Mixed Models Analysis; Mean Difference (Net) = -12.149, 95% CI 2-sided [-112.350 to 88.052] — [estimate comment as in outcome 1, analysis 1]

12. Primary Outcome: Summary of Urine 11-dehydrothromboxane B2 and Absolute Change From Baseline (ng/g) by Study Group and Visit From Week 1 to Week 24 (mITT Population) [ALCS-RA-17-11-EV]
Description: Summary of urine 11-dehydrothromboxane B2 (ng/g) and absolute change from Baseline in Weeks 12, 18 and 24 are presented (Study ALCS-RA-17-11-EV).
  The first urine void of the day was collected at Visits 1, 3 and 5 of the ALCS-RA-17-11-EV study. Baseline samples were collected Week 1 of the ALCS-RA-16-06-EV study.
  Urine creatinine concentration was measured in the urine collection and used to adjust the urine biomarker concentration value as follows:
  Urine biomarker (ng/g creatinine) = urine biomarker (pg/mL) x 100 / creatinine (mg/dL)
  Change from Baseline was calculated as follows:
  Absolute change from baseline = Post Product Use Value - Baseline Value, where Baseline = values reported on Day 1 (Week 1) of the 12-week ALCS-RA-16-06-EV study
  Baseline = Day 1 (Week 1), Visit 1 = Week 12 (Day 84 ± 3), Visit 3 = Week 18 (Day 126 ± 3), and Visit 5 = Week 24 (Day 168 ± 3), relative to the start of the 12-week ALCS-RA-16-06-EV study
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Test 1 | Test 2 | Test 1 + Test 2 Group | Control
Number analyzed (Participants) | 47 | 50 | 97 | 48
ng/g
  Baseline: Week 1 | 710.827 (429.3286) | 750.519 (463.9992) | 731.287 (445.6561) | 842.642 (493.4473)
  Visit 1: Week 12: number analyzed (Participants) | 46 | 50 | 96 | 47
  Visit 1: Week 12 | 616.618 (317.4293) | 703.961 (467.6549) | 662.109 (403.0592) | 856.055 (517.3135)
  Visit 3: Week 18: number analyzed (Participants) | 40 | 48 | 88 | 46
  Visit 3: Week 18 | 665.371 (399.2899) | 731.003 (403.6885) | 701.170 (400.7346) | 942.559 (644.6484)
  Visit 5: Week 24: number analyzed (Participants) | 42 | 48 | 90 | 43
  Visit 5: Week 24 | 567.102 (375.2503) | 706.929 (341.1676) | 641.676 (362.2939) | 969.562 (545.1937)
  Change from Baseline (Week 12): number analyzed (Participants) | 46 | 50 | 96 | 47
  Change from Baseline (Week 12) | -93.029 (372.9436) | -46.559 (438.0320) | -68.826 (406.6859) | 6.436 (462.7865)
  Change from Baseline (Week 18): number analyzed (Participants) | 40 | 48 | 88 | 46
  Change from Baseline (Week 18) | -68.815 (363.6867) | -14.677 (390.0280) | -39.285 (377.1052) | 107.568 (617.2994)
  Change from Baseline (Week 24): number analyzed (Participants) | 42 | 48 | 90 | 43
  Change from Baseline (Week 24) | -165.586 (402.1370) | -47.287 (382.6278) | -102.493 (394.1247) | 103.927 (469.7284)
Statistical Analysis 1: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0567, Mixed Models Analysis; Mean Difference (Net) = -111.957, 95% CI 2-sided [-227.151 to 3.237] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.2103, Mixed Models Analysis; Mean Difference (Net) = -76.728, 95% CI 2-sided [-197.025 to 43.569] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0052, Mixed Models Analysis; Mean Difference (Net) = -169.735, 95% CI 2-sided [-288.220 to -51.251] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.3490, Mixed Models Analysis; Mean Difference (Net) = -52.505, 95% CI 2-sided [-162.721 to 57.711] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.8410, Mixed Models Analysis; Mean Difference (Net) = -11.413, 95% CI 2-sided [-123.333 to 100.507] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.3465, Mixed Models Analysis; Mean Difference (Net) = -53.565, 95% CI 2-sided [-165.400 to 58.270] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Test 1 + Test 2 Group; Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 + Test 2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 + Test 2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 + Test 2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 + Test 2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0087, Mixed Models Analysis; Mean Difference (Net) = -111.650, 95% CI 2-sided [-194.865 to -28.435] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Control; Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Control is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Control is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Control is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Control is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.2688, Mixed Models Analysis; Mean Difference (Net) = 63.944, 95% CI 2-sided [-49.678 to 177.565] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Control; Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Control is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Control is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Control is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Control is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0096, Mixed Models Analysis; Mean Difference (Net) = 151.222, 95% CI 2-sided [37.114 to 265.330] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Control; Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Control is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Control is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Control is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Control is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0023, Mixed Models Analysis; Mean Difference (Net) = 182.631, 95% CI 2-sided [65.754 to 299.509] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.1612, Mixed Models Analysis; Mean Difference (Net) = -175.901, 95% CI 2-sided [-390.865 to 39.063] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0396, Mixed Models Analysis; Mean Difference (Net) = -227.950, 95% CI 2-sided [-448.725 to -7.175] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0002, Mixed Models Analysis; Mean Difference (Net) = -352.366, 95% CI 2-sided [-573.315 to -131.418] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.5616, Mixed Models Analysis; Mean Difference (Net) = -116.449, 95% CI 2-sided [-327.445 to 94.547] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.2176, Mixed Models Analysis; Mean Difference (Net) = -162.635, 95% CI 2-sided [-375.570 to 50.299] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0242, Mixed Models Analysis; Mean Difference (Net) = -236.196, 95% CI 2-sided [-451.334 to -21.059] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: Test 1 + Test 2 Group vs Control; Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 + Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 + Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 + Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 1 + Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -294.281, 95% CI 2-sided [-434.513 to -154.050] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: Test 1 vs Test 2; Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is NOT equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine 11-dehydrothromboxane B2 (ng/g creatinine) in Test 2 is NOT equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.1524, Mixed Models Analysis; Mean Difference (Net) = -116.170, 95% CI 2-sided [-275.521 to 43.180] — [estimate comment as in outcome 1, analysis 1]

13. Primary Outcome: Summary of Plasma sICAM-1 and Absolute Change From Baseline (ng/mL) by Study Group and Visit From Week 1 to Week 12 (mITT Population) [ALCS-RA-16-06-EV]
Description: Summary of plasma soluble Intercellular Adhesion Molecule-1 (sICAM-1) (ng/mL) and absolute change from Baseline in Weeks 6 and 12 are presented (Study ALCS-RA-16-06-EV).
  Blood samples were collected via direct venipuncture at Visits 3, 5, and 7.
  Absolute change from baseline = Post Product Use Value - Baseline Value
  Baseline / Visit 3 (Week 1) = Day 1 Visit 5 (Week 6) = Day 42 ± 3 Visit 7 (Week 12) = Day 84 ± 3
Time Frame: 12 weeks total with measurement timepoints at Week 1/Baseline, Week 6 and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Test 1 | Test 2 | Test 1 + Test 2 | Control
Number analyzed (Participants) | 127 | 131 | 258 | 139
ng/mL
  Visit 3 (Baseline): Week 1 | 230.4 (76.704) | 222.8 (77.888) | 226.6 (77.250) | 230.6 (77.084)
  Visit 5: Week 6: number analyzed (Participants) | 124 | 126 | 250 | 136
  Visit 5: Week 6 | 198.5 (54.783) | 199.8 (65.911) | 199.2 (60.529) | 224.6 (64.515)
  Visit 7: Week 12: number analyzed (Participants) | 111 | 120 | 231 | 129
  Visit 7: Week 12 | 204.1 (58.502) | 197.7 (71.517) | 200.8 (65.523) | 224.3 (70.515)
  Change from Baseline (Week 6): number analyzed (Participants) | 124 | 126 | 250 | 136
  Change from Baseline (Week 6) | -31.96 (50.532) | -22.43 (47.510) | -27.16 (49.166) | -6.613 (39.668)
  Change from Baseline (Week 12): number analyzed (Participants) | 111 | 120 | 231 | 129
  Change from Baseline (Week 12) | -23.71 (52.739) | -25.34 (46.825) | -24.56 (49.652) | -7.056 (37.619)
Statistical Analysis 1: Comparison: Test 1; Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -32.792, 95% CI 2-sided [-39.375 to -26.208] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 1; Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -25.921, 95% CI 2-sided [-33.398 to -18.443] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -25.484, 95% CI 2-sided [-31.990 to -18.979] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -26.899, 95% CI 2-sided [-34.135 to -19.663] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Test 1 + Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 + Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 + Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 + Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 + Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -26.410, 95% CI 2-sided [-31.716 to -21.103] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Control; Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Control is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Control is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Control is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Control is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p = 0.0280, Mixed Models Analysis; Mean Difference (Net) = -7.021, 95% CI 2-sided [-13.278 to -0.763] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Control; Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Control is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Control is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Control is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Control is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p = 0.0972, Mixed Models Analysis; Mean Difference (Net) = -5.902, 95% CI 2-sided [-12.881 to 1.077] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -25.771, 95% CI 2-sided [-37.189 to -14.353] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p = 0.0005, Mixed Models Analysis; Mean Difference (Net) = -20.019, 95% CI 2-sided [-32.833 to -7.205] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); p = 0.0002, Mixed Models Analysis; Mean Difference (Net) = -18.463, 95% CI 2-sided [-29.825 to -7.101] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p = 0.0002, Mixed Models Analysis; Mean Difference (Net) = -20.997, 95% CI 2-sided [-33.619 to -8.375] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Test 1 + Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 + Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 + Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 + Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 + Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -20.508, 95% CI 2-sided [-29.061 to -11.955] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Test 1 vs Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is equal to Test 2 on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to Test 2 on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is equal to Test 2 on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to Test 2 on Visit 7 (Week 12). (mITT Population); p = 0.8504, Mixed Models Analysis; Mean Difference (Net) = 0.978, 95% CI 2-sided [-9.216 to 11.172] — [estimate comment as in outcome 1, analysis 1]

14. Primary Outcome: Summary of Plasma sICAM-1 and Absolute Change From Baseline (ng/mL) by Study Group and Visit From Week 1 to Week 24 (mITT Population) [ALCS-RA-17-11-EV]
Description: Summary of plasma sICAM-1 (ng/mL) and absolute change from Baseline in Weeks 12, 18 and 24 are presented (Study ALCS-RA-17-11-EV).
  Blood samples were collected via direct venipuncture on Visits 1, 3 and 5 of the ALCS-RA-17-11-EV study. Baseline samples were collected Week 1 of the ALCS-RA-16-06-EV study.
  Change from Baseline was calculated as follows:
  Absolute change from baseline = Post Product Use Value - Baseline Value, where Baseline = values reported on Day 1 (Week 1) of the 12-week ALCS-RA-16-06-EV study
  Baseline = Day 1 (Week 1), Visit 1 = Week 12 (Day 84 ± 3), Visit 3 = Week 18 (Day 126 ± 3), and Visit 5 = Week 24 (Day 168 ± 3), relative to the start of the 12-week ALCS-RA-16-06-EV study
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Test 1 | Test 2 | Test 1 + Test 2 | Control
Number analyzed (Participants) | 47 | 50 | 97 | 49
ng/mL
  Baseline: Week 1 | 206.6 (60.303) | 205.0 (57.117) | 205.8 (58.381) | 241.3 (81.966)
  Visit 1: Week 12 | 184.0 (48.515) | 176.7 (41.375) | 180.2 (44.893) | 229.5 (69.888)
  Visit 3: Week 18: number analyzed (Participants) | 40 | 49 | 89 | 47
  Visit 3: Week 18 | 187.9 (52.027) | 182.2 (50.009) | 184.8 (50.712) | 244.9 (85.893)
  Visit 5: Week 24: number analyzed (Participants) | 42 | 47 | 89 | 44
  Visit 5: Week 24 | 184.4 (55.223) | 184.7 (62.726) | 184.6 (58.971) | 244.3 (78.272)
  Change from Baseline (Week 12) | -22.54 (45.013) | -28.33 (49.987) | -25.52 (47.484) | -11.80 (36.195)
  Change from Baseline (Week 18): number analyzed (Participants) | 40 | 49 | 89 | 47
  Change from Baseline (Week 18) | -26.73 (53.383) | -23.27 (57.191) | -24.82 (55.227) | 1.702 (47.092)
  Change from Baseline (Week 24): number analyzed (Participants) | 42 | 47 | 89 | 44
  Change from Baseline (Week 24) | -25.36 (56.800) | -21.06 (67.737) | -23.09 (62.500) | 2.091 (47.116)
Statistical Analysis 1: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 1 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 1 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -31.257, 95% CI 2-sided [-41.957 to -20.557] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 1 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 1 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -29.862, 95% CI 2-sided [-44.234 to -15.491] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 1 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 1 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -31.512, 95% CI 2-sided [-46.971 to -16.053] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 2 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 2 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -37.197, 95% CI 2-sided [-47.522 to -26.872] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 2 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 2 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -31.442, 95% CI 2-sided [-44.960 to -17.923] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0002, Mixed Models Analysis; Mean Difference (Net) = -28.597, 95% CI 2-sided [-43.340 to -13.853] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Test 1 + Test 2; Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 1 + Test 2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 + Test 2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 1 + Test 2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 + Test 2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -30.054, 95% CI 2-sided [-40.943 to -19.166] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Control; Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Control is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Control is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Control is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Control is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.2667, Mixed Models Analysis; Mean Difference (Net) = -5.904, 95% CI 2-sided [-16.370 to 4.563] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Control; Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Control is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Control is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Control is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Control is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.2085, Mixed Models Analysis; Mean Difference (Net) = 8.767, 95% CI 2-sided [-4.950 to 22.485] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Control; Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Control is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Control is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Control is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Control is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.1041, Mixed Models Analysis; Mean Difference (Net) = 12.455, 95% CI 2-sided [-2.595 to 27.505] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 1 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 1 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0058, Mixed Models Analysis; Mean Difference (Net) = -25.353, 95% CI 2-sided [-45.410 to -5.295] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 1 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 1 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0010, Mixed Models Analysis; Mean Difference (Net) = -38.630, 95% CI 2-sided [-65.062 to -12.197] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 1 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 1 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0005, Mixed Models Analysis; Mean Difference (Net) = -43.967, 95% CI 2-sided [-72.443 to -15.491] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 2 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 2 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0003, Mixed Models Analysis; Mean Difference (Net) = -31.293, 95% CI 2-sided [-51.159 to -11.428] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 2 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 2 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0004, Mixed Models Analysis; Mean Difference (Net) = -40.209, 95% CI 2-sided [-65.941 to -14.477] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0011, Mixed Models Analysis; Mean Difference (Net) = -41.052, 95% CI 2-sided [-68.965 to -13.138] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: Test 1 + Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 1 + Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 + Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 1 + Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 1 + Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -42.509, 95% CI 2-sided [-60.902 to -24.116] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: Test 1 vs Test 2; Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 2 is equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is NOT equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Plasma sICAM-1 (ng/mL) in Test 2 is equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Plasma sICAM-1 (ng/mL) in Test 2 is NOT equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.7835, Mixed Models Analysis; Mean Difference (Net) = -2.915, 95% CI 2-sided [-23.855 to 18.025] — [estimate comment as in outcome 1, analysis 1]

15. Primary Outcome: Summary of Whole Blood WBC Absolute Change From Baseline (10^3 Cells/uL) by Study Group From Week 1 to Week 12 (mITT Population With Outliers Excluded) [ALCS-RA-16-06-EV]
Description: Summary of whole blood WBC absolute change from Baseline in Week 12 is presented (Study ALCS-RA-16-06-EV).
  Blood samples were collected via direct venipuncture at Visits 3 and 7 and analyzed for the biomarker. Data outliers were examined through Proc Mixed model residual diagnosis (+/- 4 studentized residuals). A sensitivity analysis excluding outliers was performed for Visit 7 (Week 12).
  Absolute change from baseline = Post Product Use Value - Baseline Value
  Baseline / Visit 3 (Week 1) = Day 1 Visit 7 (Week 12) = Day 84 ± 3
Time Frame: Week 1 (Baseline) and Week 12 for a total of of 12 weeks from randomization
Population: Modified ITT Population with Outliers Excluded: All subjects were randomized according to the randomization schedule; who used at least one study products after randomization was recorded and for whom there was a valid (within ±3 days of the planned measurement day) baseline and at least one post-baseline biomarker. Data outliers, defined as any observation with a studentized residual that is greater than +/- 4, were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Test 1 | Test 2 | Control
Number analyzed (Participants) | 110 | 118 | 128
10^3 cells/uL | -0.564 (1.8111) | -0.389 (1.7261) | 0.227 (1.6425)
Statistical Analysis 1: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population with Outliers Excluded); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population with Outliers Excluded); p = 0.0002, Mixed Models Analysis; Mean Difference (Net) = -0.769, 95% CI 2-sided [-1.228 to -0.309] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population with Outliers Excluded); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Whole Blood WBC (x 10^3/uL) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population with Outliers Excluded); p = 0.0175, Mixed Models Analysis; Mean Difference (Net) = -0.520, 95% CI 2-sided [-0.972 to -0.068] — [estimate comment as in outcome 1, analysis 1]

16. Primary Outcome: Summary of Serum HDL-C Absolute Change From Baseline (mg/dL) by Study Group From Week 1 to Week 12 (mITT Population With Outliers Excluded) [ALCS-RA-16-06-EV]
Description: Summary of serum HDL-C absolute change from Baseline in Week 12 is presented (Study ALCS-RA-16-06-EV).
  Blood samples were collected via direct venipuncture at Visits 3 and 7 and analyzed for the biomarker. Data outliers were examined through Proc Mixed model residual diagnosis (+/- 4 studentized residuals). A sensitivity analysis excluding outliers was performed for Visit 7 (Week 12).
  Absolute change from baseline = Post Product Use Value - Baseline Value
  Baseline / Visit 3 (Week 1) = Day 1 Visit 7 (Week 12) = Day 84 ± 3
Time Frame: Week 1 (Baseline) and Week 12 for a total of of 12 weeks from randomization
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Test 1 | Test 2 | Control
Number analyzed (Participants) | 110 | 117 | 127
mg/dL | 3.3 (6.68) | 2.3 (6.95) | 0.4 (7.54)
Statistical Analysis 1: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population with Outliers Excluded); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Serum HDL-C (mg/dL) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population with Outliers Excluded); p = 0.0362, Mixed Models Analysis; Mean Difference (Net) = 2.408, 95% CI 2-sided [0.110 to 4.705] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 2 vs Control; [analysis description as in outcome 7, analysis 11]; Test type: Equivalence — [test comment as in outcome 7, analysis 11]; p = 0.2142, Mixed Models Analysis; Mean Difference (Net) = 1.692, 95% CI 2-sided [-0.569 to 3.953] — [estimate comment as in outcome 1, analysis 1]

17. Primary Outcome: Summary of Urine 8-epi-prostaglandin F2alpha Absolute Change From Baseline (ng/g) by Study Group From Week 1 to Week 12 (mITT Population With Outliers Excluded) [ALCS-RA-16-06-EV]
Description: Summary of urine 8-epi-prostaglandin F2alpha absolute change from Baseline in Week 12 is presented (Study ALCS-RA-16-06-EV).
  The first urine void of the day on Visits 3 and 7 was analyzed for the urine biomarker. Data outliers were examined through Proc Mixed model residual diagnosis (+/- 4 studentized residuals). A sensitivity analysis excluding outliers was performed for Visit 7 (Week 12).
  Urine creatinine concentration was measured in the urine collection and used to adjust the urine biomarker concentration value as follows:
  Urine biomarker (ng/g creatinine) = urine biomarker (pg/mL) x 100 / creatinine (mg/dL)
  Absolute change from baseline = Post Product Use Value - Baseline Value
  Baseline / Visit 3 (Week 1) = Day 1 Visit 7 (Week 12) = Day 84 ± 3
Time Frame: Week 1 (Baseline) and Week 12 for a total of of 12 weeks from randomization
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Test 1 | Test 2 | Control
Number analyzed (Participants) | 108 | 120 | 125
ng/g | -61.644 (138.3599) | -18.092 (135.9049) | -11.452 (133.6618)
Statistical Analysis 1: Comparison: Test 1 vs Control; [analysis description as in outcome 9, analysis 9]; Test type: Equivalence — [test comment as in outcome 9, analysis 9]; p = 0.0250, Mixed Models Analysis; Mean Difference (Net) = -39.501, 95% CI 2-sided [-75.396 to -3.605] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 2 vs Control; [analysis description as in outcome 9, analysis 11]; Test type: Equivalence — [test comment as in outcome 9, analysis 11]; p = 0.9997, Mixed Models Analysis; Mean Difference (Net) = -2.940, 95% CI 2-sided [-37.896 to 32.016] — [estimate comment as in outcome 1, analysis 1]

18. Primary Outcome: Summary of Urine 11-dehydrothromboxane B2 Absolute Change From Baseline (ng/g) by Study Group From Week 1 to Week 12 (mITT Population With Outliers Excluded) [ALCS-RA-16-06-EV]
Description: Summary of urine 11-dehydrothromboxane B2 absolute change from Baseline in Week 12 is presented (Study ALCS-RA-16-06-EV).
  The first urine void of the day on Visits 3 and 7 was analyzed for the urine biomarker. Data outliers were examined through Proc Mixed model residual diagnosis (+/- 4 studentized residuals). A sensitivity analysis excluding outliers was performed for Visit 7 (Week 12).
  Urine creatinine concentration was measured in the urine collection and used to adjust the urine biomarker concentration value as follows:
  Urine biomarker (ng/g creatinine) = urine biomarker (pg/mL) x 100 / creatinine (mg/dL)
  Absolute change from baseline = Post Product Use Value - Baseline Value
  Baseline / Visit 3 (Week 1) = Day 1 Visit 7 (Week 12) = Day 84 ± 3
Time Frame: Week 1 (Baseline) and Week 12 for a total of of 12 weeks from randomization
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Test 1 | Test 2 | Control
Number analyzed (Participants) | 110 | 120 | 124
ng/g | -47.736 (488.1213) | -55.751 (486.6897) | -3.878 (414.5263)
Statistical Analysis 1: Comparison: Test 1 vs Control; [analysis description as in outcome 11, analysis 9]; Test type: Equivalence — [test comment as in outcome 11, analysis 9]; p = 0.6778, Mixed Models Analysis; Mean Difference (Net) = -54.398, 95% CI 2-sided [-177.281 to 68.485] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 2 vs Control; [analysis description as in outcome 11, analysis 11]; Test type: Equivalence — [test comment as in outcome 11, analysis 11]; p = 0.7497, Mixed Models Analysis; Mean Difference (Net) = -48.395, 95% CI 2-sided [-168.697 to 71.908] — [estimate comment as in outcome 1, analysis 1]

19. Primary Outcome: Summary of Plasma sICAM-1 Absolute Change From Baseline (ng/mL) by Study Group From Week 1 to Week 12 (mITT Population With Outliers Excluded) [ALCS-RA-16-06-EV]
Description: Summary of plasma sICAM-1 absolute change from Baseline in Week 12 is presented (Study ALCS-RA-16-06-EV).
  Blood samples were collected via direct venipuncture at Visits 3 and 7 and analyzed for the biomarker. Data outliers were examined through Proc Mixed model residual diagnosis (+/- 4 studentized residuals). A sensitivity analysis excluding outliers was performed for Visit 7 (Week 12).
  Absolute change from baseline = Post Product Use Value - Baseline Value
  Baseline / Visit 3 (Week 1) = Day 1 Visit 7 (Week 12) = Day 84 ± 3
Time Frame: Week 1 (Baseline) and Week 12 for a total of of 12 weeks from randomization
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Test 1 | Test 2 | Control
Number analyzed (Participants) | 111 | 119 | 129
ng/mL | -23.71 (52.739) | -26.02 (46.433) | -7.056 (37.619)
Statistical Analysis 1: Comparison: Test 1 vs Control; [analysis description as in outcome 13, analysis 9]; Test type: Equivalence — [test comment as in outcome 13, analysis 9]; p = 0.0003, Mixed Models Analysis; Mean Difference (Net) = -20.010, 95% CI 2-sided [-32.447 to -7.573] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 2 vs Control; [analysis description as in outcome 13, analysis 11]; Test type: Equivalence — [test comment as in outcome 13, analysis 11]; p < .0001, Mixed Models Analysis; Mean Difference (Net) = -22.566, 95% CI 2-sided [-34.837 to -10.295] — [estimate comment as in outcome 1, analysis 1]

20. Primary Outcome: Summary of Urine Total NNAL Absolute Change From Baseline (ng/g) by Study Group From Week 1 to Week 12 (mITT Population With Outliers Excluded) [ALCS-RA-16-06-EV]
Description: Summary of urine total NNAL absolute change from Baseline in Week 12 is presented (Study ALCS-RA-16-06-EV).
  The first urine void of the day on Visits 3 and 7 was analyzed for the urine biomarker. Data outliers were examined through Proc Mixed model residual diagnosis (+/- 4 studentized residuals). A sensitivity analysis excluding outliers was performed for Visit 7 (Week 12).
  Urine creatinine concentration was measured in the urine collection and used to adjust the urine biomarker concentration value as follows:
  Urine biomarker (ng/g creatinine) = urine biomarker (pg/mL) x 100 / creatinine (mg/dL)
  Absolute change from baseline = Post Product Use Value - Baseline Value
  Baseline / Visit 3 (Week 1) = Day 1 Visit 7 (Week 12) = Day 84 ± 3
Time Frame: Week 1 (Baseline) and Week 12 for a total of of 12 weeks from randomization
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Test 1 | Test 2 | Control
Number analyzed (Participants) | 112 | 120 | 128
ng/g | -191.327 (220.6982) | -160.201 (192.1456) | -15.898 (149.1447)
Statistical Analysis 1: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -179.365, 95% CI 2-sided [-225.708 to -133.022] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Total NNAL (ng/g creatinine) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p < .0001, Mixed Models Analysis; Mean Difference (Net) = -153.220, 95% CI 2-sided [-198.930 to -107.509] — [estimate comment as in outcome 1, analysis 1]

21. Primary Outcome: Summary of Whole Blood COHB Absolute Change From Baseline (% Saturation) by Study Group From Week 1 to Week 12 (mITT Population With Outliers Excluded) [ALCS-RA-16-06-EV]
Description: Summary of whole blood COHB absolute change from Baseline in Week 12 is presented (Study ALCS-RA-16-06-EV).
  Blood samples were collected via direct venipuncture at Visits 3 and 7 and analyzed for the biomarker. Data outliers were examined through Proc Mixed model residual diagnosis (+/- 4 studentized residuals). A sensitivity analysis excluding outliers was performed for Visit 7 (Week 12).
  Absolute change from baseline = Post Product Use Value - Baseline Value
  Baseline / Visit 3 (Week 1) = Day 1 Visit 7 (Week 12) = Day 84 ± 3
Time Frame: Week 1 (Baseline) and Week 12 for a total of of 12 weeks from randomization
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Test 1 | Test 2 | Control
Number analyzed (Participants) | 110 | 120 | 128
percent saturation | -2.57 (2.363) | -2.44 (2.187) | 0.07 (1.920)
Statistical Analysis 1: Comparison: Test 1 vs Control; [analysis description as in outcome 3, analysis 9]; Test type: Equivalence — [test comment as in outcome 3, analysis 9]; p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.569, 95% CI 2-sided [-3.084 to -2.054] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 2 vs Control; [analysis description as in outcome 3, analysis 11]; Test type: Equivalence — [test comment as in outcome 3, analysis 11]; p < .0001, Mixed Models Analysis; Mean Difference (Net) = -2.586, 95% CI 2-sided [-3.092 to -2.081] — [estimate comment as in outcome 1, analysis 1]

22. Secondary Outcome: Frequency of eCO as Compliance Indicator, Weeks 12 (Study ALCS-RA-16-06-EV) and 24 (Study ALCS-RA-17-11-EV)
Description: Participant compliance for the abstention of any type of tobacco/nicotine product for the duration of the study was assessed by measuring the participant's exhaled carbon monoxide (eCO, ppm). According to their eCO measurements at Weeks 12 (study ALCS-RA-16-06-EV) and Week 24 (study ALCS-RA-17-11-EV), participants were categorized into 1 of 3 categories: 'eCO ≤ 5', 'eCO < 5 - ≤ 8', or 'eCO > 8'. Lower eCO values represent lower smoking exposure and increased compliance, with the 'eCO ≤ 5' category indicating that the participant abstained from smoking, the 'eCO < 5 - ≤ 8' category indicating low smoking exposure to the participant, and the 'eCO > 8' category indicating non-compliance with the study criteria that the participant refrain from smoking during the study.
Time Frame: Weeks 12 (Study ALCS-RA-16-06-EV) and Week 24 (Study ALCS-RA-17-11-EV) from randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Test 1 | Test 2
Number analyzed (Participants) | 112 | 121
Participants
  Exhaled CO at Week 12: eCO ≤ 5 | 76 | 77
  Exhaled CO at Week 12: eCO < 5 - ≤ 8 | 13 | 21
  Exhaled CO at Week 12: eCO > 8 | 23 | 23
  Exhaled CO at Week 24: number analyzed (Participants) | 42 | 48
  Exhaled CO at Week 24: eCO ≤ 5 | 35 | 40
  Exhaled CO at Week 24: eCO < 5 - ≤ 8 | 5 | 4
  Exhaled CO at Week 24: eCO > 8 | 2 | 4

23. Secondary Outcome: Percentage of Predicted FEV1 and Absolute Change From Baseline to Week 12 by Study Group (mITT Population) [ALCS-RA-16-06-EV]
Description: Percentage of predicted forced expiratory volume in the first second (FEV1) and absolute change from Baseline to Week 12 by Study Group is presented (Study ALCS-RA-16-06-EV).
  Baseline / Screening = Day -28 to Day -5 Visit 7 (Week 12) = Day 84 ± 3
  Absolute change from baseline = Post Product Use Value - Baseline Value
  FEV1 = Forced Expiratory Volume in 1 Second
Time Frame: Assessments at Screening (Day -28 to Day -5) and Week 12 (Day 84 +/- 3 )
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Test 1 | Test 2 | Test 1 + Test 2 Group | Control
Number analyzed (Participants) | 100 | 112 | 212 | 115
percentage of predicted FEV1
  Screening (Baseline) | 91.059 (13.9979) | 91.335 (12.8396) | 91.205 (13.3671) | 90.139 (13.4146)
  Week 12 | 89.989 (13.7140) | 90.918 (13.3174) | 90.480 (13.4818) | 87.743 (13.4729)
  Change from Baseline at Week 12 | -1.070 (6.5798) | -0.416 (5.4848) | -0.725 (6.0205) | -2.396 (6.2471)
Statistical Analysis 1: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FEV1 (%) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FEV1 (%) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FEV1 (%) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FEV1 (%) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p = 0.0839, ANCOVA; Mean Difference (Net) = 1.42, 95% CI 2-sided [-0.19 to 3.04] — The ANCOVA includes study group, gender, and age class as fixed effects, and baseline score as the covariate. Least-squares means (LS Means) are calculated from the ANCOVA
Statistical Analysis 2: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FEV1 (%) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FEV1 (%) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FEV1 (%) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FEV1 (%) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p = 0.0089, ANCOVA; Mean Difference (Net) = 2.10, 95% CI 2-sided [0.53 to 3.66] — [estimate comment as in outcome 23, analysis 1]

24. Secondary Outcome: Percentage of Predicted FVC and Absolute Change From Baseline to Week 12 by Study Group (mITT Population) [ALCS-RA-16-06-EV]
Description: Percentage of predicted forced vital capacity (FVC) and absolute change from Baseline to Week 12 by Study Group is presented (Study ALCS-RA-16-06-EV).
  Baseline / Screening = Day -28 to Day -5 Visit 7 (Week 12) = Day 84 ± 3
  Absolute change from baseline = Post Product Use Value - Baseline Value
  FVC = Forced Vital Capacity
Time Frame: Assessments at Screening (Day -28 to Day -5) and Week 12 (Day 84 +/- 3 )
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of predicted FVC
Arm/Group | Test 1 | Test 2 | Test 1 + Test 2 Group | Control
Number analyzed (Participants) | 100 | 112 | 212 | 115
percentage of predicted FVC
  Screening (Baseline) | 92.709 (12.7747) | 93.789 (11.7222) | 93.280 (12.2126) | 92.809 (12.2784)
  Week 12 | 91.733 (13.3234) | 92.730 (11.9222) | 92.260 (12.5822) | 91.552 (12.7403)
  Change from Baseline at Week 12 | -0.976 (5.1281) | -1.059 (5.3244) | -1.020 (5.2205) | -1.257 (5.1665)
Statistical Analysis 1: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FVC (%) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FVC (%) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FVC (%) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FVC (%) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p = 0.7101, ANCOVA; Mean Difference (Net) = 0.26, 95% CI 2-sided [-1.13 to 1.66] — [estimate comment as in outcome 23, analysis 1]
Statistical Analysis 2: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FVC (%) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FVC (%) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FVC (%) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FVC (%) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p = 0.7325, ANCOVA; Mean Difference (Net) = 0.24, 95% CI 2-sided [-1.12 to 1.59] — [estimate comment as in outcome 23, analysis 1]

25. Secondary Outcome: Percentage of Predicted FEV1/FVC and Absolute Change From Baseline to Week 12 by Study Group (mITT Population) [ALCS-RA-16-06-EV]
Description: Percentage of predicted FEV1/FVC and absolute change from Baseline to Week 12 by Study Group is presented (Study ALCS-RA-16-06-EV).
  Baseline / Screening = Day -28 to Day -5 Visit 7 (Week 12) = Day 84 ± 3
  Absolute change from baseline = Post Product Use Value - Baseline Value
  FEV1 = Forced Expiratory Volume in 1 Second, FVC = Forced Vital Capacity.
Time Frame: Assessments at Screening (Day -28 to Day -5) and Week 12 (Day 84 +/- 3 )
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1/FVC
Arm/Group | Test 1 | Test 2 | Test 1 + Test 2 Group | Control
Number analyzed (Participants) | 100 | 112 | 212 | 115
percentage of predicted FEV1/FVC
  Screening (Baseline) | 98.202 (7.5989) | 97.535 (7.9699) | 97.849 (7.7859) | 97.243 (8.1131)
  Week 12 | 98.219 (7.7279) | 98.135 (7.3706) | 98.175 (7.5234) | 95.959 (8.1492)
  Change from Baseline at Week 12 | 0.017 (4.4796) | 0.600 (3.3508) | 0.325 (3.9251) | -1.285 (5.5994)
Statistical Analysis 1: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FEV1/FVC (%) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FEV1/FVC (%) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FEV1/FVC (%) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FEV1/FVC (%) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p = 0.0136, ANCOVA; Mean Difference (Net) = 1.48, 95% CI 2-sided [0.31 to 2.66] — [estimate comment as in outcome 23, analysis 1]
Statistical Analysis 2: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FEV1/FVC (%) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FEV1/FVC (%) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FEV1/FVC (%) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Screening) for Percentage of Predicted FEV1/FVC (%) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p = 0.0009, ANCOVA; Mean Difference (Net) = 1.94, 95% CI 2-sided [0.80 to 3.08] — [estimate comment as in outcome 23, analysis 1]

26. Other Pre Specified Outcome: Summary of Urine Nicotine Equivalents and Absolute Change From Baseline (mg/g) by Study Group and Visit From Week 1 to Week 12 (mITT Population) [ALCS-RA-16-06-EV]
Description: Summary of urine Nicotine Equivalents (mg/g) and absolute change from Baseline in Weeks 6 and 12 are presented (Study ALCS-RA-16-06-EV).
  The first urine void of the day was collected at Visits 3, 5 and 7.
  Nicotine equivalents (μg/mL) = (nicotine [ng/mL]/162.23 [mg/mmol] + nicotinegluc (ng/mL)/338.36 [mg/mmol] + cotinine [ng/mL]/176.22 [mg/mmol] + cotininegluc [ng/mL]/352.34 [mg/mmol] + trans-3'-hydroxycotinine [ng/mL]/192.22 [mg/mmol] + trans-3'-hydroxycotinine-gluc [ng/mL]/368.34 [mg/mmol]) x 162.23 (mg/mmol) x 1 μg/1000 ng
  Urine creatinine concentration was measured in the urine collection and used to adjust the urine biomarker concentration value as follows:
  Urine biomarker (ng/g creatinine) = urine biomarker (pg/mL) x 100 / creatinine (mg/dL)
  Absolute change from baseline = Post Product Use Value - Baseline Value
  Baseline / Visit 3 (Week 1) = Day 1 Visit 5 (Week 6) = Day 42 ± 3 Visit 7 (Week 12) = Day 84 ± 3
Time Frame: 12 weeks total with measurement timepoints at Week 1/Baseline, Week 6 and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Test 1 | Test 2 | Test 1 + Test 2 | Control
Number analyzed (Participants) | 127 | 131 | 258 | 138
mg/g
  Visit 3 (Baseline): Week 1 | 10.865 (5.6124) | 10.629 (5.5776) | 10.745 (5.5851) | 11.126 (5.5647)
  Visit 5: Week 6: number analyzed (Participants) | 124 | 123 | 247 | 134
  Visit 5: Week 6 | 10.666 (7.4649) | 10.026 (7.0465) | 10.347 (7.2519) | 10.766 (5.3662)
  Visit 7: Week 12: number analyzed (Participants) | 112 | 119 | 231 | 127
  Visit 7: Week 12 | 10.869 (7.5555) | 11.054 (7.0353) | 10.965 (7.2768) | 10.268 (5.5748)
  Change from Baseline (Week 6): number analyzed (Participants) | 124 | 123 | 247 | 134
  Change from Baseline (Week 6) | -0.109 (5.7252) | -0.600 (5.0695) | -0.353 (5.4032) | -0.499 (3.4735)
  Change from Baseline (Week 12): number analyzed (Participants) | 112 | 119 | 231 | 127
  Change from Baseline (Week 12) | 0.219 (5.2922) | 0.435 (4.9935) | 0.330 (5.1304) | -0.943 (3.4975)
Statistical Analysis 1: Comparison: Test 1; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p = 0.9294, Mixed Models Analysis; Mean Difference (Net) = 0.038, 95% CI 2-sided [-0.795 to 0.870] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 1; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p = 0.5290, Mixed Models Analysis; Mean Difference (Net) = 0.277, 95% CI 2-sided [-0.587 to 1.142] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p = 0.2291, Mixed Models Analysis; Mean Difference (Net) = -0.508, 95% CI 2-sided [-1.337 to 0.321] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p = 0.2179, Mixed Models Analysis; Mean Difference (Net) = 0.525, 95% CI 2-sided [-0.311 to 1.361] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Test 1 + Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 + Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 + Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 + Test 2 is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 + Test 2 is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p = 0.2002, Mixed Models Analysis; Mean Difference (Net) = 0.401, 95% CI 2-sided [-0.213 to 1.016] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Control is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Control is NOT equal to zero on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Control is equal to zero on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Control is NOT equal to zero on Visit 5 (Week 6). (mITT Population); p = 0.4760, Mixed Models Analysis; Mean Difference (Net) = -0.290, 95% CI 2-sided [-1.089 to 0.509] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Control is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Control is NOT equal to zero on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Control is equal to zero on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Control is NOT equal to zero on Visit 7 (Week 12). (mITT Population); p = 0.0914, Mixed Models Analysis; Mean Difference (Net) = -0.699, 95% CI 2-sided [-1.512 to 0.113] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); p = 0.9705, Mixed Models Analysis; Mean Difference (Net) = 0.328, 95% CI 2-sided [-1.122 to 1.777] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p = 0.3280, Mixed Models Analysis; Mean Difference (Net) = 0.977, 95% CI 2-sided [-0.512 to 2.465] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is equal to Control on Visit 5 (Week 6). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is NOT equal to Control on Visit 5 (Week 6). (mITT Population); p = 0.9951, Mixed Models Analysis; Mean Difference (Net) = -0.218, 95% CI 2-sided [-1.667 to 1.230] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p = 0.1367, Mixed Models Analysis; Mean Difference (Net) = 1.225, 95% CI 2-sided [-0.244 to 2.693] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Test 1 + Test 2 vs Control; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 + Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 + Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 + Test 2 is equal to Control on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 + Test 2 is NOT equal to Control on Visit 7 (Week 12). (mITT Population); p = 0.0294, Mixed Models Analysis; Mean Difference (Net) = 1.101, 95% CI 2-sided [0.111 to 2.091] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Test 1 vs Test 2; Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to Test 2 on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to Test 2 on Visit 7 (Week 12). (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to Test 2 on Visit 7 (Week 12). Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to Test 2 on Visit 7 (Week 12). (mITT Population); p = 0.6792, Mixed Models Analysis; Mean Difference (Net) = -0.248, 95% CI 2-sided [-1.424 to 0.928] — [estimate comment as in outcome 1, analysis 1]

27. Other Pre Specified Outcome: Summary of Urine Nicotine Equivalents and Absolute Change From Baseline (mg/g) by Study Group and Visit From Week 1 to Week 24 (mITT Population) [ALCS-RA-17-11-EV]
Description: Summary of urine nicotine equivalents (mg/g Cr) and absolute change from Baseline in Weeks 12, 18 and 24 are presented (Study ALCS-RA-17-11-EV).
  The first urine void of the day was collected at Visits 1, 3 and 5 of the ALCS-RA-17-11-EV study. Baseline samples were collected Week 1 of the ALCS-RA-16-06-EV study.
  Nicotine equivalents (μg/mL) = (nicotine [ng/mL]/162.23 [mg/mmol] + nicotinegluc (ng/mL)/338.36 [mg/mmol] + cotinine [ng/mL]/176.22 [mg/mmol] + cotininegluc [ng/mL]/352.34 [mg/mmol] + trans-3'-hydroxycotinine [ng/mL]/192.22 [mg/mmol] + trans-3'-hydroxycotinine-gluc [ng/mL]/368.34 [mg/mmol]) x 162.23 (mg/mmol) x 1 μg/1000 ng
  Urine creatinine concentration was measured in the urine collection and used to adjust the urine biomarker concentration value as follows:
  Urine biomarker (ng/g creatinine) = urine biomarker (pg/mL) x 100 / creatinine (mg/dL)
  Change from Baseline was calculated as follows:
  Absolute change from baseline = Post Product Use Value - Baseline Val
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Test 1 | Test 2 | Test 1 + Test 2 Group | Control
Number analyzed (Participants) | 47 | 50 | 97 | 49
mg/g
  Baseline: Week 1 | 10.107 (4.9952) | 10.684 (5.2636) | 10.404 (5.1168) | 11.813 (5.4517)
  Visit 1: Week 12 | 10.412 (7.7828) | 11.949 (7.0536) | 11.205 (7.4173) | 11.101 (5.7563)
  Visit 3: Week 18: number analyzed (Participants) | 40 | 48 | 88 | 47
  Visit 3: Week 18 | 12.421 (9.6385) | 11.634 (7.8863) | 11.992 (8.6833) | 10.841 (5.4127)
  Visit 5: Week 24: number analyzed (Participants) | 42 | 48 | 90 | 44
  Visit 5: Week 24 | 10.621 (8.5013) | 12.782 (7.1436) | 11.773 (7.8370) | 10.442 (4.5456)
  Change from Baseline (Week 12) | 0.305 (5.4615) | 1.266 (5.5160) | 0.800 (5.4823) | -0.713 (3.9573)
  Change from Baseline (Week 18): number analyzed (Participants) | 40 | 48 | 88 | 47
  Change from Baseline (Week 18) | 2.360 (6.9077) | 1.281 (6.3017) | 1.771 (6.5677) | -0.976 (4.4242)
  Change from Baseline (Week 24): number analyzed (Participants) | 42 | 48 | 90 | 44
  Change from Baseline (Week 24) | 0.680 (5.9020) | 2.103 (7.0107) | 1.439 (6.5202) | -1.372 (4.1783)
Statistical Analysis 1: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.4012, Mixed Models Analysis; Mean Difference (Net) = 0.638, 95% CI 2-sided [-0.860 to 2.137] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0201, Mixed Models Analysis; Mean Difference (Net) = 2.163, 95% CI 2-sided [0.343 to 3.983] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test 1; Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.1709, Mixed Models Analysis; Mean Difference (Net) = 1.210, 95% CI 2-sided [-0.528 to 2.948] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0307, Mixed Models Analysis; Mean Difference (Net) = 1.593, 95% CI 2-sided [0.150 to 3.035] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0691, Mixed Models Analysis; Mean Difference (Net) = 1.588, 95% CI 2-sided [-0.126 to 3.302] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Test 2; Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0034, Mixed Models Analysis; Mean Difference (Net) = 2.487, 95% CI 2-sided [0.838 to 4.137] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Test 1 + Test 2 Group; Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 + Test 2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 + Test 2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 + Test 2 is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 + Test 2 is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0034, Mixed Models Analysis; Mean Difference (Net) = 1.849, 95% CI 2-sided [0.622 to 3.075] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Control; Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Control is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Control is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Control is equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Control is NOT equal to zero on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.8123, Mixed Models Analysis; Mean Difference (Net) = -0.178, 95% CI 2-sided [-1.654 to 1.299] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Control; Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Control is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Control is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Control is equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Control is NOT equal to zero on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.5879, Mixed Models Analysis; Mean Difference (Net) = -0.480, 95% CI 2-sided [-2.226 to 1.267] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Control; Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Control is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Control is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Control is equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Control is NOT equal to zero on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.4910, Mixed Models Analysis; Mean Difference (Net) = -0.596, 95% CI 2-sided [-2.304 to 1.111] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.9673, Mixed Models Analysis; Mean Difference (Net) = 0.816, 95% CI 2-sided [-1.967 to 3.599] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.1787, Mixed Models Analysis; Mean Difference (Net) = 2.643, 95% CI 2-sided [-0.683 to 5.968] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Test 1 vs Control; Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.5243, Mixed Models Analysis; Mean Difference (Net) = 1.806, 95% CI 2-sided [-1.406 to 5.018] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is NOT equal to Control on Visit 1 (Week 12), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.3956, Mixed Models Analysis; Mean Difference (Net) = 1.770, 95% CI 2-sided [-0.966 to 4.507] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is NOT equal to Control on Visit 3 (Week 18), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.3810, Mixed Models Analysis; Mean Difference (Net) = 2.068, 95% CI 2-sided [-1.160 to 5.295] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Test 2 vs Control; Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0557, Mixed Models Analysis; Mean Difference (Net) = 3.084, 95% CI 2-sided [-0.049 to 6.216] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: Test 1 + Test 2 Group vs Control; Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 + Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 + Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 + Test 2 is equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 1 + Test 2 is NOT equal to Control on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.0195, Mixed Models Analysis; Mean Difference (Net) = 2.445, 95% CI 2-sided [0.400 to 4.490] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: Test 1 vs Test 2; Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is NOT equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); Test type: Equivalence — Null hypothesis: Absolute change from Baseline for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. Alternate hypothesis: Absolute change from Baseline (Week 1) for Urine Nicotine Equivalents (mg/g creatinine) in Test 2 is NOT equal to Test 1 on Visit 5 (Week 24), relative to the start of the 12-week ALCS-RA-16-06-EV study. (mITT Population); p = 0.2817, Mixed Models Analysis; Mean Difference (Net) = -1.277, 95% CI 2-sided [-3.615 to 1.060] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and recorded from the time of Screening/Visit 2 of the 12-week ALCS-RA-16-06-EV study until Week 24/ End of Study of the ALCS-RA-17-11-EV extension study (or upon early termination).
Description: After completing screening at Visit 2 of the ALCS-RA-16-06-EV study, eligible subjects were randomized to a study group. Eligible subjects completing ALCS-RA-16-06-EV were enrolled in the ALCS-RA-17-11-EV extension study to the same study group. Adverse events are reported per study (ALCS-RA-16-06-EV or ALCS-RA-17-11-EV).
Groups:
- Test 1 (ALCS-RA-16-06-EV): Subjects were instructed to stop use of their own brand of cigarettes and were provided with exclusive ad libitum use of e-vapor Test Product 1 (Nu Mark LLC, MarkTen® XL Bold CLASSIC*) without use of any other type of tobacco/nicotine containing product, for the entire duration of participation in study ALCS-RA-16-06-EV.
  *Product no longer sold commercially
- Test 2 (ALCS-RA-16-06-EV): Subjects were instructed to stop use of their own brand of cigarettes and were provided with exclusive ad libitum use of e-vapor Test Product 2 (Nu Mark LLC, MarkTen® XL Bold MENTHOL*) without use of any other type of tobacco/nicotine containing product, for the entire duration of participation in study ALCS-RA-16-06-EV.
  *Product no longer sold commercially
- Control (ALCS-RA-16-06-EV): Subjects continued smoking their own brand of conventional lit-end cigarettes under ad libitum use of, without use of any other type of tobacco/nicotine containing product, for the entire duration of participation in study ALCS-RA-16-06-EV.
- Overall (ALCS-RA-16-06-EV): This group consists of all subjects who participated in study ALCS-RA-16-06-EV and were assigned to the Test 1 group, the Test 2 group or the Control group.
- Test 1 (ALCS-RA-17-11-EV): Subjects were instructed to stop use of their own brand of cigarettes and were provided with exclusive ad libitum use of e-vapor Test Product 1 (Nu Mark LLC, MarkTen® XL Bold CLASSIC*) without use of any other type of tobacco/nicotine containing product, for the entire duration of participation in study ALCS-RA-17-11-EV.
  *Product no longer sold commercially
- Test 2 (ALCS-RA-17-11-EV): Subjects were instructed to stop use of their own brand of cigarettes and were provided with exclusive ad libitum use of e-vapor Test Product 2 (Nu Mark LLC, MarkTen® XL Bold MENTHOL*) without use of any other type of tobacco/nicotine containing product, for the entire duration of participation in study ALCS-RA-17-11-EV.
  *Product no longer sold commercially
- Control (ALCS-RA-17-11-EV): Subjects continued smoking their own brand of conventional lit-end cigarettes under ad libitum use of, without use of any other type of tobacco/nicotine containing product, for the entire duration of participation in study ALCS-RA-17-11-EV.
- Overall (ALCS-RA-17-11-EV): This group consists of all subjects who participated in study ALCS-RA-17-11-EV and were assigned to the Test 1 group, the Test 2 group or the Control group.
Arm/Group | Test 1 (ALCS-RA-16-06-EV) | Test 2 (ALCS-RA-16-06-EV) | Control (ALCS-RA-16-06-EV) | Overall (ALCS-RA-16-06-EV) | Test 1 (ALCS-RA-17-11-EV) | Test 2 (ALCS-RA-17-11-EV) | Control (ALCS-RA-17-11-EV) | Overall (ALCS-RA-17-11-EV)
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/150 | 0/149 | 0/450 | 0/48 | 0/50 | 0/52 | 0/150
Serious Adverse Events (participants affected / at risk) | 1/151 | 1/150 | 1/149 | 3/450 | 0/48 | 0/50 | 0/52 | 0/150
Other Adverse Events (participants affected / at risk) | 49/151 | 47/150 | 24/149 | 120/450 | 13/48 | 15/50 | 10/52 | 38/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test 1 (ALCS-RA-16-06-EV) (N=151) | Test 2 (ALCS-RA-16-06-EV) (N=150) | Control (ALCS-RA-16-06-EV) (N=149) | Overall (ALCS-RA-16-06-EV) (N=450) | Test 1 (ALCS-RA-17-11-EV) (N=48) | Test 2 (ALCS-RA-17-11-EV) (N=50) | Control (ALCS-RA-17-11-EV) (N=52) | Overall (ALCS-RA-17-11-EV) (N=150)
Multiple fractures secondary to motor vehicle accident (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Subject 5048 had multiple fractures due to a road traffic accident during Week 8 of the study. The subject completed the study. The PI considered the multiple fractures, road traffic accident, and hematoma (on scalp) not related to study product.
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Subject 9082 experienced suicidal ideation during Week 8 of study. Subject failed to report his history of treatment for psychiatric condition since age 16. The PI considered suicidal ideation unlikely to be related, or not related, to the product.
MISCARRIAGE (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Subject 6105 was found to be pregnant during Week 12 of the study and was discontinued. On 18 July 2017, the subject reported that she had a spontaneous miscarriage at home the day prior. The PI considered this event not related to study product.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test 1 (ALCS-RA-16-06-EV) (N=151) | Test 2 (ALCS-RA-16-06-EV) (N=150) | Control (ALCS-RA-16-06-EV) (N=149) | Overall (ALCS-RA-16-06-EV) (N=450) | Test 1 (ALCS-RA-17-11-EV) (N=48) | Test 2 (ALCS-RA-17-11-EV) (N=50) | Control (ALCS-RA-17-11-EV) (N=52) | Overall (ALCS-RA-17-11-EV) (N=150)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemoconcentration (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteogenesis imperfecta (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroglossal cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 4 (4) | 0 (0) | 7 (7) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival recession (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Multiple allergies (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abscess jaw (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asymptomatic bacteriuria (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 3 (8) | 0 (0) | 8 (14) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fractured coccyx (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 2 (4) | 1 (1) | 4 (6) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 2 (3)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bilirubin urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonoscopy (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematocrit increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine ketone body present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urobilinogen urine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food craving (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Muscle strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (6) | 3 (3) | 2 (2) | 10 (11) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 2 (3)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7) | 1 (1) | 13 (13) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0) | 6 (6) | 1 (1) | 2 (3) | 0 (0) | 3 (4)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (7):
  • Study Protocol: ALCS-RA-16-06-EV Protocol Version 1 (2016-11-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT04800211/Prot_000.pdf
  • Study Protocol: ALCS-RA-16-06-EV Protocol Version 2 (2016-12-07): https://cdn.clinicaltrials.gov/large-docs/11/NCT04800211/Prot_001.pdf
  • Study Protocol: ALCS-RA-17-11-EV Protocol Version 1 (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT04800211/Prot_002.pdf
  • Study Protocol: ALCS-RA-17-11-EV Protocol Version 2 (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT04800211/Prot_003.pdf
  • Study Protocol: ALCS-RA-17-11-EV Protocol Version 3 (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/11/NCT04800211/Prot_004.pdf
  • Statistical Analysis Plan: ALCS-RA-16-06-EV Statistical Analysis Plan Version 1 (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/11/NCT04800211/SAP_005.pdf
  • Statistical Analysis Plan: ALCS-RA-17-11-EV Statistical Analysis Plan Version 1 (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT04800211/SAP_006.pdf